

# NCT03600805

# STATISTICAL ANALYSIS PLAN

A randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of sarilumab in patients with giant cell arteritis

#### SAR153191-EFC15068

| STATISTICIAN: | | |
|----------------------------|------------------------|----|
| DATE OF ISSUE: 08-Jan-2021 | | |
| | Total number of pages: | 87 |

Any and all information presented in this document shall be treated as confidential and shall remain the exclusive property of Sanofi (or any of its affiliated companies). The use of such confidential information must be restricted to the recipient for the agreed purpose and must not be disclosed, published or otherwise communicated to any unauthorized persons, for any reason, in any form whatsoever without the prior written consent of Sanofi (or the concerned affiliated company); 'affiliated company' means any corporation, partnership or other entity which at the date of communication or afterwards (i) controls directly or indirectly Sanofi, (ii) is directly or indirectly controlled by Sanofi, with 'control' meaning direct or indirect ownership of more than 50% of the capital stock or the voting rights in such corporation, partnership or other entity

According to template: QSD-002643 VERSION 6.0 (06-JUL-2016)

# **TABLE OF CONTENTS**

| STATIS | TICAL ANALYSIS PLAN | 1 |
|---|---|---|
| TABLE | OF CONTENTS | 2 |
| LIST OF | F ABBREVIATIONS AND DEFINITION OF TERMS | 5 |
| 1 | OVERVIEW AND INVESTIGATIONAL PLAN | |
| 1.1 | STUDY DESIGN AND RANDOMIZATION | |
| 1.1 | | |
| 1.2 | OBJECTIVES | |
| 1.2.1 | Primary objectives | 8 |
| 1.2.2 | Secondary objectives | 8 |
| 1.2.3 | Other objectives | 8 |
| 1.3 | DETERMINATION OF SAMPLE SIZE | 9 |
| 1.4 | STUDY PLAN | 10 |
| 1.5 | MODIFICATIONS TO THE STATISTICAL SECTION OF THE PROTOCOL | 12 |
| 1.6 | STATISTICAL MODIFICATIONS MADE IN THE STATISTICAL ANALYSIS PLAN | 12 |
| 2 | STATISTICAL AND ANALYTICAL PROCEDURES | 14 |
| 2.1 | ANALYSIS ENDPOINTS | 14 |
| 2.1.1 | Demographic and baseline characteristics | 14 |
| 2.1.2 | Prior or concomitant medications | 16 |
| 2.1.3 | Efficacy endpoints | 16 |
| 2.1.3.1 | Primary efficacy endpoint(s) | 16 |
| 2.1.3.2 | Secondary efficacy endpoint(s) | 19 |
| 2.1.4 | Safety endpoints | |
| 2.1.4.1 | Adverse events variables | |
| 2.1.4.2<br>2.1.4.3 | Deaths | |
| 2.1.4.3 | Vital signs variables | |
| 2.1.4.5 | Antinuclear antibodies | |
| 2.1.5 | Immunogenicity endpoints | 27 |
| 2.1.6 | Pharmacokinetic variables | 28 |
| 2.1.7 | Pharmacodynamic/genomics endpoints | 28 |
| 218 | Other efficacy endpoints | 28 |

| 4 | DATABASE LOCK | 53 |
|---|---|---|
| 3 | INTERIM ANALYSIS | 52 |
| 2.5.8 | Statistical technical issues | 51 |
| 2.5.7 | Pooling of centers for statistical analyses | 51 |
| 2.5.6 | Remote Assessment | 50 |
| 2.5.5 | Unscheduled visits | 50 |
| 2.5.4 | Windows for time points | 50 |
| 2.5.3 | Missing data | 49 |
| 2.5.2 | Data handling conventions for secondary efficacy variables | 48 |
| 2.5.1 | General conventions | 48 |
| 2.5 | DATA HANDLING CONVENTIONS | 48 |
| 2.4.9 | DNA/RNA | 48 |
| 2.4.8 | Analysis of immunogenicity endpoints | 47 |
| 2.4.7 | Analyses of quality of life variables | 46 |
| 2.4.6 | Analyses of pharmacokinetic variables | 46 |
| 2.4.5.4 | Analyses of laboratory variables | |
| 2.4.5.2<br>2.4.5.3 | Deaths Analyses of laboratory variables | |
| 2.4.5.1 | Analyses of adverse events | 42 |
| 2.4.5 | Analyses of safety data | |
| 2.4.4.2<br>2.4.4.3 | Analyses of secondary efficacy endpoints | |
| 2.4.4.1 | Analysis of primary and additional efficacy endpoint(s) | |
| 2.4.4 | Analyses of efficacy endpoints | 38 |
| 2.4.3.2 | Compliance | |
| 2.4.3<br>2.4.3.1 | Extent of investigational medicinal product exposure and compliance Extent of investigational medicinal product exposure | |
| 2.4.2 | Prior or concomitant medications. | |
| 2.4.1 | Demographics and baseline characteristics | |
| 2.4 | STATISTICAL METHODS | |
| 2.3.3 | Pharmacokinetics and ADA populations | 36 |
| 2.3.2 | Safety population | |
| 2.3.1<br>2.3.1.1 | Efficacy populations Intent-to-treat population | 35 |
| 2.3 | ANALYSIS POPULATIONS | |
| 2.2.1 | Randomization and drug dispensing irregularities | |
| 2.2 | DISPOSITION OF PATIENTS | |

| 5 S | SOFTWARE DOCUMENTATION | . 54 |
|---|---|---|
| 6 R | REFERENCES | . 55 |
| 7 L | IST OF APPENDICES | .56 |
| APPENDIX | K A STUDY FLOW CHART | .57 |
| APPENDIX | K B POTENTIALLY CLINICALLY SIGNIFICANT ABNORMALITIES (PCSA) CRITERIA | .62 |
| APPENDIX | C SUMMARY OF STATISTICAL ANALYSES | .68 |
| APPENDIX | K D SF-36 V2 SCORING | .71 |
| APPENDIX | K E FACIT-FATIGUE SCORING GUIDELINES (VERSION 4) | .73 |
| APPENDIX | K F SAS CODE FOR EQ-5D-3L INDEX UTILITY SCORING | .74 |
| APPENDIX | K G SAS CODE FOR SF-36 SCORING | .75 |
| APPENDIX | K H VISIT WINDOWS BASED ON DAY RANGES | .83 |
| APPENDIX | K L. BASELINE GLUCOCORTICOID TOXICITY | 86 |

# LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

ADA: antidrug antibody AEs: adverse events

AESIs: adverse events of special interest

ALP: alkaline phosphatase
ALT: alanine aminotransferase
ANA: antinuclear antibodies
AST: asparate aminotransferase

BMI: body mass index
CRF: case report form
CSR: clinical study report
ds-DNA: double-stranded DNA

EOS: end of study

EQ-5D-3L: EuroQol five-dimensional three-level questionnaire

FACIT-Fatigue: functional assessment of chronic illness therapy fatigue scale

GTI: glucocorticoid toxicity index

HAQ-DI: health assessment questionnaire disability index

HbA1c: hemoglobin A1c

HDL-C: high density lipoprotein cholesterol

HLGT: high level group term HLT: high level term

ID: identification

IMP: investigational medicinal product

LDH: lactate dehydrogenase

LDL-C: low density lipoprotein cholesterol

LLN: lower limit of normal

LLOQ: lower limit of quantification

LLT: lower level term

MD-VAS: physician global assessment of disease activity- visual analog scale

MedDRA: Medical Dictionary for Regulatory Activities

NCEP ATPIII: National Cholesterol Education Program Adult Treatment Panel III

PRO: patient reported outcome

PT: preferred term RBC: red blood cell

SAEs: serious adverse events SF-36v2: short form 36 version 2 SOC: system organ class

TEAE: treatment-emergent adverse event

ULN: upper limit of normal WBC: white blood cell

WHO-DD: World Health Organization - Drug Dictionary

# 1 OVERVIEW AND INVESTIGATIONAL PLAN

This statistical analysis plan (SAP) provides a comprehensive and detailed description of statistical strategy and methodology to be used to analyze the data from sarilumab EFC15068 study in patients with giant cell arteritis (GCA).

Due to the ongoing pandemic of COVID-19 (the disease caused by the novel coronavirus), the operations of sarilumab (Kevzara®) clinical trial EFC15068 have been significantly disrupted in various countries and sites. Consequently, the screening/recruitment activities for this study have been suspended since 19<sup>th</sup> of March 2020. Due to the protracted recruitment timeline and internal portfolio reprioritization, in July 2020, Sanofi has decided not to re-open the screening/recruitment activities and to discontinue the study. This decision is not related to any safety issues arising from the administration of sarilumab.

A total of 83 patients (out of 360 planned patients) have been randomized in the study. While the number of randomized patients may not be adequate to demonstrate a statistically significant benefit, the data generated from the treated patients may contribute to the further understanding of IL-6 signaling blockade in this disease state.

## 1.1 STUDY DESIGN AND RANDOMIZATION

#### Original study design

This is a multicenter, randomized, double-blind, placebo controlled 52-week Phase 3 study with a 24-week post-treatment follow up phase, evaluating the efficacy and safety of sarilumab in patients with giant cell arteritis (GCA).

Approximately 360 patients with GCA (new onset or refractory [eg, disease relapse] GCA) who meet the entry criteria will be randomized to 4 parallel treatment groups with sarilumab 200 mg q2w, 150 mg q2w, or placebo q2w plus 26-week prednisone taper, or placebo q2w with 52-week standardized prednisone taper at a ratio of 2:1:1:2 as described below. Randomization will be stratified by the starting dose of prednisone at baseline (<30 mg/day or  $\ge$ 30 mg/day) using a block randomization schedule, and aim to enroll at least 30% of new onset patients by capping enrolment of refractory patients to  $\le$ 70% of total patients randomized.

- Treatment Group A: sarilumab 200 mg q2w with a 26-week taper of CS.
- Treatment Group B: sarilumab 150 mg q2w with a 26-week taper of CS.
- Treatment Group C: sarilumab matching placebo q2w with a 26-week taper of CS.
- Treatment Group D: sarilumab matching placebo q2w with a 52-week taper of CS.

It is important to optimize CS treatment prior to randomization to minimize the risk of adverse sequelae from GCA. Patients will be dosed with prednisone between 20 to 60 mg/day at the time of randomization (baseline) and initiate a taper according to the protocol defined schedule. Patients will be initiated on a standardized taper of prednisone from the time of randomization.

The taper will initially be open label; patients will have between 1 to 7 weeks to taper prednisone dose to 20 mg/day following randomization.

The further tapering of prednisone once a dose of 20 mg/day is achieved will be done in a blinded manner. To achieve the appropriate daily dose during this phase, patients will receive a combination of prednisone and/or placebo to prednisone depending on the assigned treatment group and associated taper regimen.

The total tapering period (open label plus double blind prednisone periods) will be between 46 weeks to 52 weeks depending on the initial prednisone dose at randomization.

At each site visit, the patient's disease will be assessed to determine whether the patient can adhere to the protocol defined prednisone taper schedule.

During the course of study, for patients in need of rescue therapy as per Investigator judgment, CS should be the agent of first choice. Patients may continue SC administration of sarilumab or matching placebo only if CS is used as the rescue therapy. If the patients remain symptomatic despite CS rescue therapy, then other treatment options including nonbiological immunosuppressive drugs may be used and the patient must be discontinued from the study treatment and considered a non-responder.

If the patient or Investigator decides to discontinue the administration of blinded sarilumab injections, then the patient will be asked to return to the site for study assessments as per protocol until end of study (EOS) evaluation, unless the patient cannot or does not wish to continue the assessments, in which case an early withdrawal visit and safety follow up should be performed. It is recommended that patients complete Visit 13, if possible.

Total duration of study participation for each patient is up to 82 weeks:

- Up to 6 weeks screening period.
- 52-week treatment period (sarilumab or placebo, double-blind phase).
- 24-week post treatment follow-up period.

The last patient last visit will occur when the last patient has completed the 24-week follow up period (EOS). The end of the clinical trial is defined as the last patient's last visit.

## Study discontinuation plan

As mentioned in Section 1, due to the protracted recruitment timeline and internal portfolio reprioritization, Sanofi has decided to terminate the EFC15068 study in July 2020. For patients who were already enrolled with ongoing treatment in the study, investigators were instructed to discontinue the study drugs and transition these patients into post-treatment follow-up period for safety assessments. The study discontinuation plan is as follows:

• All randomized patients should stop by 12 weeks from the date of announcement to the sites and should be scheduled for the end of study treatment visit at their earliest

convenience and no later than *October 13, 2020*, which would ensure sufficient time for patients to identify alternative therapy as needed.

• All patients will have a follow-up (EOS) visit that is 6 weeks after treatment cessation and no later than *November 24, 2020*.

Thus, the last patient last visit will occur when the last patient has completed the 6-week follow-up period (EOS). The end of the clinical trial is defined as the last patient's last visit.

#### 1.2 OBJECTIVES

## 1.2.1 Primary objectives

To evaluate the efficacy of sarilumab in patients with GCA as assessed by the proportion of patients with sustained remission at Week 52 for sarilumab compared to placebo, in combination with a 26-week CS tapering course.

## 1.2.2 Secondary objectives

- To demonstrate the efficacy of sarilumab in patients with GCA compared to placebo, in combination with (either 26 or 52 weeks) CS tapering course with regard to:
  - Clinical responses (such as responses based on disease remission rates, time to first disease flare) over time.
  - Cumulative CS (including prednisone) exposure.
- To assess the safety (including immunogenicity) and tolerability of sarilumab in patients with GCA.
- To measure sarilumab serum concentrations in patients with GCA.
- To assess the effect of sarilumab on sparing glucocorticoid toxicity as measured by glucocorticoid toxicity index (GTI).

#### 1.2.3 Other objectives

- To assess the effect of sarilumab on physician assessment of disease activity as measured by a visual analogue scale (MD-VAS).
- To assess the effect of sarilumab compared with placebo, in combination with a 26-week CS taper as on a variety of patient reported outcome (PRO) concepts including fatigue (FACIT-Fatigue), health status (EuroQol five-dimensional three-level questionnaire [EQ-5D-3L], Short form 36 version 2 [SF-36v2]), physical functioning (health assessment questionnaire disability index [HAQ-DI]), including pain (visual analogue scale) and patient assessment of disease activity (visual analogue scale).
- To assess the impact of ESR/CRP levels on remission status.

- To characterize the disease activity of GCA patients while on steroid taper or sarilumab treatment in a subset of patients using comprehensive approaches to evaluate circulating immune cell types.
- To characterize the disease activity of GCA patients while on steroid taper or sarilumab treatment by evaluating circulating proteins, genetics and gene expression in consenting patients.

#### 1.3 DETERMINATION OF SAMPLE SIZE

The sample size calculations are based on the primary efficacy variable of sustained remission at Week 52. Data from another trial that evaluated the safety and efficacy of tocilizumab in a similar population show that the expected event rate in Group C (placebo with 26-week taper, n = 60) is 14% and in Group D (placebo with 52-week taper, n = 120) is 18% (1). Assuming a treatment difference of 40% and a significance level of 0.01 (2-sided) this will ensure that all comparisons of the primary endpoint in Group A (sarilumab 200 mg, n = 120) and Group B (sarilumab 150 mg, n = 60) compared to the 2 control groups will have at least 90% power. The sample size has also been selected to ensure adequate power for sensitivity analyses excluding acute phase reactants from the primary endpoint definition.

The above calculations were for the full enrollment. However, the number of randomized patients is 83 in 4 arms at the time of the premature termination of the study. In addition, based on patients' enrollment dates and the study discontinuation plan, only about 36 patients (out of 83) had an opportunity to complete the 52-week treatment period. For the cohort of patients who did not have an opportunity to complete the 52-week treatment period, it is not meaningful to define the endpoint of sustained remission at Week 52. Therefore, the analysis of primary endpoint will be limited to the cohort of patients who had an opportunity to complete the 52-week treatment period. Due to the small number of patients (n=36) in this cohort (see Section 2.3.1 for definition of the cohort), the powers on the primary endpoint are minimal. As a result, all the efficacy analyses will be descriptive in nature and all reported p-values will be nominal for the study.

Based on patients' enrollment dates, all enrolled patients (n=83) had an opportunity to complete at least 24 weeks of treatment, therefore, an additional endpoint, sustained remission at Week 24 is added in the SAP (see Section 2.1.3.1 for the detail definition). Table 1 provides the power calculations on the additional endpoint of sustained remission at Week 24. Due to the small number of patients in each individual treatment group, the power calculations were also provided for the comparison between the combined sarilumab groups (i.e., Group A+B) and the combined placebo groups (i.e., Group C+D) assuming the same effect sizes as mentioned above.

Table 1: Updated power calculations

| | Estimate of | |
|-----------|---------------|-----------|
| | the sustained | Estimated |
| | remission | Sample |
| Treatment | rate | size |
| Group A | 54% | 28 |
| Group B | 50% | 14 |

| | Power [1] | Power [2] |
|------------------------|-----------|-----------|
| 6 | | |
| Comparison | (%) | (%) |
| Group A versus Group C | 45.7 | 74.0 |
| Group A versus Group D | 58.6 | 81.1 |

| 08-Jan-2021 | |
|-----------------|---|
| Version number: | 1 |

| Group C | 14% | 14 |
|-----------------------------------|-----|----|
| Group D | 18% | 27 |
| Group A + B (combined sarilumab) | 53% | 42 |
| Group C + D<br>(combined placebo) | 17% | 41 |

| Group B versus Group C | 28.1 | 53.5 |
|---|---|---|
| Group B versus Group D | 33.6 | 57.1 |
| Group A+B versus Group<br>C+D | 82.3 | 94.5 |
| Power [1] was based on an alpha level of 0.01.<br>Power [2] was based on an alpha level of 0.05. | | |

Treatment Group A: sarilumab 200 mg q2w with a 26 week taper of CS.

Treatment Group B: sarilumab 150 mg q2w with a 26 week taper of CS.

Treatment Group C: sarilumab matching placebo q2w with a 26 week taper of CS.

Treatment Group D: sarilumab matching placebo q2w with a 52 week taper of CS.

Powers were calculated using the Chi-square test for each comparison; Calculations were made using nQuery Advisor 7.0.

#### 1.4 STUDY PLAN

The schedule of the safety, efficacy, pharmacokinetic (PK), and immunogenicity assessments from Section 1.2 of the study protocol is provided in Appendix A. The graphical study design is provided in Figure 1.

08-Jan-2021 Version number: 1

Figure 1 - Graphic study design



Patients will be randomized to 4 groups with the ratio of 2:1:1:2

\*Patients experiencing a disease flare may be rescued with open-label treatment as per Investigator judgment during the study treatment period.

#### 1.5 MODIFICATIONS TO THE STATISTICAL SECTION OF THE PROTOCOL

There was one protocol amendment for EFC15068 study (see Table 2). The overall rationale for the changes implemented in the protocol amendment 01 was to address several comments raised by the European Regulatory Authorities during the initial protocol review. The changes made in the statistical section in the protocol amendment 01 are summarized in Table 3.

Table 2: Protocol amendment history

| Document | Country/Countries impacted by amendement | Date, version |
|---|---|---|
| Amended Clinical Trial Protocol 01 | All | 12-Sep-2018, version 1 (electronic 2.0) |
| Original Protocol | All | 09-Feb-2018, version 1 (electronic 4.0) |

Table 3: Summary of changes of the statistical section - Protocol amendment 01

| Section # and<br>Name | Description of Change | Brief Rationale |
|---|---|---|
| Clinical Trial Summary –Statistical Consideration AND Section 11.1 Determination of sample size | More details on the power calculations were added. | The assumed treatment effects used for the power calculations were added for clarity. |
| Section 11.4.2.1<br>Analysis of primary<br>efficacy endpoint(s) | The non-inferiority test between Sarilumab 200 mg q2w arm and the placebo with 52 weeks taper arm was removed. | Based on the results from the GiACTA study, the non-<br>inferiority test is deemed as unnecessary and thus<br>removed from the protocol |
| Section 11.4.2.3<br>Multiplicity<br>considerations | The hierarchical testing approach including the testing sequence for the secondary endpoints were clarified. | Details on the hierarchical testing sequence for the secondary endpoints were added for clarification to address a specific request from the European Regulatory Authorities. |

## 1.6 STATISTICAL MODIFICATIONS MADE IN THE STATISTICAL ANALYSIS PLAN

Due to the early termination of the study and study discontinuation plan, a large amount of data will not be able to be collected since many enrolled patients will not complete all planned study visits and study procedures for the assessments of efficacy, ADA, and biomarker endpoints. In addition, the number of randomized patients is 83 in 4 arms (out of 360 planned) at the time of the premature termination of the study. The changes from the statistical analysis plan outlined in the protocol are summarized below.

• The primary endpoint for the study is sustained remission at Week 52. Based on patients' enrollment dates and the study discontinuation plan, only about 36 patients (out of 83) had an opportunity to complete the 52-week treatment period. For the cohort of patients who

did not have an opportunity to complete the 52-week treatment period, it is not meaningful to define the endpoint of sustained remission at Week 52. Therefore, the analysis of primary endpoint will be limited to the cohort of patients who had an opportunity to complete the 52-week treatment period. Details can be found in Section 2.1.3.1 and Section 2.4.4.1.

- Based on patients' enrollment dates and the study discontinuation plan, all patients should have had the opportunity to be treated for at least 24 weeks, so an additional endpoint, sustained remission at Week 24, is added in the SAP. Details can be found in Section 2.1.3.1.
- Due to the same reason as mentioned above, the secondary endpoints of cumulative GTI scores at Week 52 will be limited to the cohort of patients who had an opportunity to complete the 52-week treatment period. In addition, the cumulative GTI scores will also be assessed at Week 24. Details are provided in Section 2.1.3.2.
- The missing data imputation strategy for defining the endpoints of sustained remission at W24 and W52, and cumulative GTI scores at W24 and W52 can be found in Section 2.1.3.1 and Section 2.1.3.2, respectively; the rest of efficacy analyses will be based on data as observed, no missing data will be imputed.
- A statistically significance level of 0.01 (2-sided) was prespecified in the protocol for all the between group comparisons. Due to reason mentioned in the first bullet, the analysis of the primary endpoint of sustained remission at Week 52 will be limited to the cohort of patients who had an opportunity to complete the 52-week treatment period (n=36). With a total of 36 patients, the powers on the primary endpoint are minimal. Therefore, all the analyses will be descriptive in nature.
  - a) For majority of the efficacy endpoints, only descriptive summary statistics will be provided by 4 treatment groups.
  - b) For the primary and some selected important secondary endpoints, summary statistics and formal statistical tests on between group comparisons (with 95% CI and p-value) will be provided for the 2 combined treatment groups (ie, 2 sarilumab groups combined versus 2 placebo groups combined). Details are provided in Section 2.4.4.
- No multiplicity/hierarchy testing will be applied; all p-values will be nominal.
- No subgroup analyses will be planned due to the small sample sizes.

# 2 STATISTICAL AND ANALYTICAL PROCEDURES

Data analyses will be performed in the double-blind (DB) 52-week treatment period. The analysis results will be presented by 4 treatment groups (Groups A, B, C and D) in the DB assessment period. The posttreatment follow-up phase will be presented separately without formal statistical testing as needed.

#### 2.1 ANALYSIS ENDPOINTS

# 2.1.1 Demographic and baseline characteristics

The baseline value is defined as the last available value prior to the first dose of study medication, SC IMP.

All baseline safety and efficacy parameters (apart from those listed below) are presented along with the on-treatment summary statistics in the efficacy and safety sections (Section 2.4.4 and Section 2.4.5).

#### Demographic characteristics

The following demographic characteristics will be summarized separately by treatment and overall:

- Sex (Male, Female)
- Race (Caucasian/White, Black, Asian/Oriental, Other)
- Ethnicity (Hispanic, Not Hispanic)
- Region (Region 1 [Western countries], Region 2 [South America], and Region 3 [Rest of the World]); definitions of the regions are provided in Section 2.5.7
- Age (years)
- Age group ( $\ge$ 50 and <65,  $\ge$ 65 and <75,  $\ge$ 75 and <85,  $\ge$ 85 years)
- Weight (kg)
- Weight group ( $<60, \ge 60 \text{ and } <100, \ge 100 \text{ kg}$ )
- Body mass index (BMI, kg/m<sup>2</sup>)
- BMI group (<25,  $\ge 25$  and <30,  $\ge 30$  kg/m<sup>2</sup>)
- Smoking status (never, former, current)
- Alcohol habits (never, occasional, monthly, weekly, daily)

## Medical or surgical history

Medical or surgical history includes all the relevant findings within the lifetime of the patient.

This information will be coded to a "Lower Level Term (LLT)", "Preferred Term (PT)", "High Level Term (HLT)", "High Level Group Term (HLGT)", and associated primary "System Organ Class (SOC)" using the version of Medical Dictionary for Regulatory Activities (MedDRA) currently in effect at Sanofi at the time of database lock.

#### Disease characteristics at baseline

The following baseline disease characteristics as well as the other baseline characteristics will be summarized separately by treatment group:

- Unequivocal cranial symptoms of GCA (Yes, No)
- Unequivocal symptoms of PMR (Yes, No)
- Other features judged by the investigator to be consistent with GCA or PMR flares (Yes, No)
- Diagnostic temporal artery biopsy (Yes, No)
- Diagnostic imaging performed (Yes, No) and imaging methodology (Angiography, CTA, MRA, PET-CT, Ultrasound)
- Duration of GCA (from diagnosis date to baseline)
- GCA Disease onset (new onset, refractory)
- Prior GCA flares (≤6 months, 6 to 12 months or >12 months prior to screening)
- Prednisone dose at baseline
- Prednisone dose group at baseline (≤30 mg/day, >30 mg/day)
- Highest dose and duration of corticosteroid taper taken for GCA within 24 weeks prior to screening
- Physician global assessment of disease activity (MD-VAS)
- C-reactive protein (CRP) at baseline
- CRP group (≤median, >median)
- ESR at baseline
- ESR group (≤median, >median)
- ESR  $\geq$  30 mm/h and/or CRP  $\geq$  10mg within 6 weeks prior to screening (Yes, No)
- Glucocorticoid toxicity at baseline\*

Any technical details related to computation, dates, and imputations for missing dates are described in Section 2.5.

<sup>\*</sup>The baseline glucocorticoid toxicity is established by a composite index calculated from weighted scores assigned by toxicities. The scores are described in Appendix I.

#### 2.1.2 Prior or concomitant medications

All medications taken within a certain period of time before randomization and until the end of the study, including vaccines taken before screening, biological/non-biological disease modifying anti-rheumatic drugs [DMARDs] and immunosuppressive agents taken for patients with symptomatic GCA disease are to be reported in the case report form (CRF) pages. The highest dose and duration of all corticosteroids taper taken for GCA within the 24 weeks prior to screening and all corticosteroids taken during the study are also reported.

All medications will be coded using the World Health Organization – Drug Dictionary (WHO-DD) version currently in effect at Sanofi at the time of database lock.

- Prior medications are those the patient used prior to first investigational medicinal product (IMP) intake. Prior medications can be discontinued before first dosing or can be ongoing during treatment phase.
- Concomitant medications are any treatments received by the patient concomitantly to the IMP, during the treatment-emergent period (Section 2.1.3).

A given medication can be classified as a prior medication, as a concomitant medication, and/or as a post-treatment medication.

For patients who experience a disease flare and are in need of rescue therapy, study patients prescribed with rescue corticosteroids (non-investigational medicinal product) per investigator judgement during the course of the study will continue administration of subcutaneous (SC) IMP (sarilumab or its matching placebo) for the full duration of the 52-week treatment period.

Any technical details related to computation, dates, imputation for missing dates are described in Section 2.5.

# 2.1.3 Efficacy endpoints

#### 2.1.3.1 Primary efficacy endpoint(s)

The primary endpoint is the proportion of patients achieving sustained remission at Week 52, where the sustained remission at Week 52 is defined as having met all following parameters:

- 1. Achievement of disease remission not later than Week 12,
- 2. Absence of disease flare from Week 12 through Week 52,
- 3. Normalization of CRP (to <10 mg/L, with an absence of successive elevations to ≥10 mg/L) from Week 12 through Week 52, and
- 4. Successful adherence to the prednisone taper from Week 12 through Week 52.

Based on patients' enrollment dates and the study discontinuation plan, not all the patients had an opportunity to complete the 52-week treatment period. For the cohort of patients who did not have an opportunity to complete the 52-week treatment period, it is not meaningful to define the endpoint of sustained remission at Week 52. Therefore, the analysis of primary endpoint will be

limited to the cohort of patients who had an opportunity to complete the 52-week treatment period. The detail definition of this cohort can be found in Section 2.3.1.

## Components of primary endpoint are described as below:

#### 1. Achievement of disease remission not later than Week 12

**Disease remission** is defined as resolution of signs and symptoms of GCA, and normalization of CRP (<10 mg/L). Note that a single CRP elevation ( $\ge10 \text{ mg/L}$ ) is not considered absence of remission unless CRP remained elevated ( $\ge10 \text{ mg/L}$ ) at the next study visit.

The status of normalization of CRP (<10 mg/L) will be determined based on the last two non-missing post-baseline CRP values measured up to Week 12. If at least one of them is <10 mg/L, then it is considered as normalization of CRP.

# Signs and symptoms of disease

Evaluation of clinical signs and symptoms by the Efficacy Assessor at every study visit according to the schedule of assessment will include the following:

- Symptoms of PMR as indicated by the Efficacy Assessor (morning stiffness and/or pain, in the shoulder and/or hip girdles)
- Cranial symptoms.
  - Localized headache.
  - Temporal artery or scalp tenderness.
  - Visual signs or symptoms such as acute or subacute vision loss due to arteritic anterior ischemic optic neuropathy (A-AION), transient blurry vision (generally monocular or at least affecting 1 eye at a time, but potentially affecting both eyes), diplopia.
  - Jaw or mouth pain, tongue claudication.
- Constitutional syndrome, including but not limited to fever, malaise, unintentional weight loss, night sweat, asthenia, fatigue, loss of appetite.
- New or worsened extremity claudication, bruits and asymmetrical pulses.
- Other features judged by the Investigator to be consistent with a GCA or PMR flare.

The resolution of signs and symptoms of GCA is identified in eCRF "GCA Assessment" page with the question "Based upon the patient's relevant medical history and the clinical assessment and responses provided above, does the patient have active GCA?" ticked as "No". The resolution of signs and symptoms of GCA by Week 12 will be determined based on the last non-missing post-baseline GCA assessment measured up to Week 12.

Patients who took rescue CS due to active GCA prior to Week 12 or who permanently withdraw from the study treatment prior to Week 12 will be considered as not achieved disease remission by Week 12.

# 2. Absence of disease flare from Week 12 through Week 52.

Flare is defined as either 1) recurrence of signs and symptoms attributable to active GCA plus an increase in CS dose due to GCA, or 2) elevation of ESR attributable to active GCA plus an increase in CS dose due to GCA. Increase in CS dose is defined as:

- Any dose increase during the protocol defined steroid taper, or
- Reinitiation of prednisone therapy after the protocol defined taper has been completed.

Patients with disease flare are identified as those with the reason for treatment ticked "rescue therapy" in eCRF "Steroid Medication" page and to the question "If Rescue Therapy, please specify" ticked either "Active GCA" or "Elevated ESR Attributable to Active GCA".

# 3. Normalization of CRP (to <10 mg/L, with an absence of successive elevations to ≥10 mg/L) from Week 12 through Week 52

The status of normalization of CRP from Week 12 through Week 52 will be determined based on the CRP values measured at Week 16, Week 20, Week 24, Week 32, Week 40 and Week 52. If there are two or more consecutive visits with CRP≥10 mg/L, then it is categorized as no normalization of CRP. Intermittent missing CRP at Week 16, Week 20, Week 24, Week 32, Week 40 or Week 52 will be imputed using last value carried forward (LOCF) approach.

#### 4. Successful adherence to the prednisone taper from Week 12 through Week 52

Successful adherence to the prednisone taper from Week 12 through Week 52 is defined as patients did not take rescue therapy from Week 12 through Week 52 and may include the use of any excess prednisone (beyond the per protocol CS tapering regimen) with a cumulative dose of ≤100 mg (or equivalent), such as those employed to manage AE not related to GCA. The cumulative dose of excess prednisone use will be counted from baseline to Week 52.

In addition, patients who permanently withdraw from the study treatment prior to Week 52 will be considered as not achieved component 2, 3, or 4 for the primary endpoint.

#### Additional Endpoint: Sustained remission at Week 24

Based on patients' enrollment dates and the study discontinuation plan, all patients would have had the opportunity to be treated for at least 24 weeks. As a result, an additional endpoint, sustained remission at Week 24, which is defined similarly as the primary endpoint but with shorter sustained period, is added in the SAP.

The sustained remission at Week 24 is defined by having met all of the following parameters:

- Achievement of disease remission not later than Week 12,
- Absence of disease flare from Week 12 through Week 24,
- Normalization of CRP (to <10 mg/L, with an absence of successive elevations to ≥10 mg/L) from Week 12 through Week 24, and
- Successful adherence to the prednisone taper from Week 12 through Week 24.

## Components of the sustained remission at Week 24 are described as below:

- 1. Achievement of disease remission not later than Week 12, which is defined in the same way as described for the primary endpoint.
- 2. Absence of disease flare from Week 12 through Week 24, where disease flare is defined in the same way as described for the primary endpoint.
- 3. Normalization of CRP (to <10 mg/L, with an absence of successive elevations to ≥10 mg/L) from Week 12 through Week 24

The status of normalization of CRP from Week 12 through Week 24 will be determined based on the CRP values measured at Week 16, Week 20, Week 24. If there are two or more consecutive visits with CRP≥10 mg/L, then it's categorized as no normalization of CRP. Intermittent missing CRP at Week 16, Week 20 or Week 24 will be imputed using last value carried forward (LOCF) approach.

# 4. Successful adherence to the prednisone taper from Week 12 through Week 24

Successful adherence to the prednisone taper from Week 12 through Week 24 is defined as patients did not take rescue therapy from Week 12 through Week 24 and may include the use of any excess prednisone (beyond the per protocol CS tapering regimen) with a cumulative dose of ≤100 mg (or equivalent), such as those employed to manage AE not related to GCA. The cumulative dose of excess prednisone use will be counted from baseline to Week 24.

In addition, patients who permanently withdraw from the study treatment prior to Week 24 will be considered as not achieved component 2, 3, or 4 for the primary endpoint.

# Blinding of CRP and ESR assessment results

Investigators, including Efficacy Assessors, and patients will remain blinded to CRP and ESR results (except screening and baseline). Safety Assessors will also be blinded on post baseline CRP but will have access to ESR results.

ESR kits will be provided by the central laboratory while the test will be performed locally at site, results (the distance in millimeters (mm) that red blood cells has descended in 1 hour) will be blinded to Investigators including Efficacy Assessors and staff directly involved in efficacy assessment of study patients.

#### 2.1.3.2 Secondary efficacy endpoint(s)

The following efficacy variables will be assessed:

- Components of sustained remission composite measure at Week 52 and Week 24
- Total cumulative corticosteroid (including prednisone) dose over during the treatment period
- Time to first GCA flare during the treatment period

• GTI Cumulative worsening score (CWS) and Aggregate improvement score (AIS) at Week 52 and Week 24.

Below are descriptions of these variables. Details related to imputation of GTI scores are described in Section 2.5.2.

# Components of sustained remission composite measure at Week 52

- 1. Proportion of patients who achieved disease remission by Week 12.
- 2. Proportion of patients who have no disease flare from Week 12 through Week 52.
- 3. Proportion of patients who have normalization of CRP (to <10 mg/L, with an absence of successive elevations to  $\ge10$  mg/L) from Week 12 through Week 52.
- 4. Proportion of patients who successfully adhere to the prednisone taper from Week 12 through Week 52.

## Components of sustained remission composite measure at Week 24

- 1. Proportion of patients who achieved disease remission by Week 12.
- 2. Proportion of patients who have no disease flare from Week 12 through Week 24.
- 3. Proportion of patients who have normalization of CRP (to <10 mg/L, with an absence of successive elevations to  $\ge10 \text{ mg/L}$ ) from Week 12 through Week 24.
- 4. Proportion of patients who successfully adhere to the prednisone taper from Week 12 through Week 24.

## Total cumulative corticosteroid (including prednisone) dose during the treatment period

The total cumulative corticosteroid includes prednisone taper regimen per protocol, use of prednisone (an excess of  $\leq 100$  mg of prednisone during the study treatment period such as those employed to manage AE not related to GCA is permissible for meeting the definition of maintenance of sustained remission) and rescue corticosteroids dose prescribed for rescue therapy over the treatment period for GCA disease only.

#### Time to first GCA flare during the treatment period

The duration (in days) from randomization to first GCA flare after clinical remission and up to 52 weeks. Patients who never achieve remission will be censored at randomization day; and those who achieved clinical remission and never flared will be censored at the end of treatment assessment date up to Week 52.

The definition of GCA flare is provide in Section 2.1.3.1 primary efficacy endpoint.

Clinical remission is defined as resolution of signs and symptoms and normalization of CRP (<10 mg/L). Intermittent missing CRP at visit will be imputed using last value carried forward (LOCF) approach. If missing signs and symptoms, then clinical remission is not achieved.

# Glucocorticoid toxicity index (GTI) scores and components

The GTI is intended to capture glucocorticoid (GC)-related morbidity and GC-sparing ability of other therapies (2).

The GTI is composed of two components, the Composite GTI and the Specific List (Table 4). The Composite GTI consists of nine domains (body mass index (BMI), glucose tolerance, blood pressure, Hyperlipidemia, Bone Health (BMD), steroid myopathy, Skin steroid-related Toxicity, Neuropsychiatric - steroid related symptoms and infection) on common steroid-related adverse events anticipated to occur in ≥5% of patients treated in a clinical trial involving glucocorticoids. The Specific List consists of 23 items (11 domains) that are mainly less common but serious adverse effects, serving as a complementary tool to the Composite GTI to ensure that all important elements of glucocorticoid toxicity were captured.

The domains of the Composite GTI and the specific list of the GTI will be assessed at baseline, Week 12, Week 24, Week 40 and Week 52, except for bone density (BMD) which will be assessed at Baseline and Week 52 only.

Please note, due to early termination of the study, most patients will not have BMD assessed at Week 52. In addition, for patients who withdraw from the study prior to Week 24, the BMD will not be measured at the EOT visit as no substantial changes are expected within 6 months of treatment. As a result, missing BMD score will be imputed as 'no change'. The BMD measured at the end of treatment (EOT) visit will be included in the definition of cumulative GTI scores (i.e., CWS and AIS as defined below) at Week 52 regardless when the EOT visit is occurred. The BMD domain score will be set to 'no change' in the calculation of the cumulative GTI scores at Week 24.

# Scoring of the Glucocorticoid Toxicity Index (GTI)

**Domain-specific score** for each patient at a visit is defined as the weight assigned based on the change in severity level as described for each domain in Table 4.

**Composite GTI score** for each patient at a visit is the sum of 9 domain-specific scores at each visit.

**Cumulative GTI score** is the sum of composite GTI score across visits. Two cumulative GTI scores, CWS and AIS, will be defined.

## • Cumulative worsening score (CWS)

CWS is designed to assess cumulative GC toxicity, regardless of whether the toxicity has lasting effects or is transient. New toxicities that occur are added, but toxicities that appear to resolve on follow-up are not removed. Thus, the CWS serves as a lasting record of GC toxicity observed and can only increase or remain the same over time.

CWS will be lower in the treatment arm compared to the placebo arm at the end of trial, if the treatment is effective at decreasing GC toxicity over time.

## • Aggregate improvement score (AIS)

Patients are anticipated to have some GC toxicity at baseline, the AIS would be important in establishing that the new therapy is effective at diminishing any baseline GC toxicity over time. With the AIS, toxicities can be removed if improvement occurs, and added if worsening occurs.

AIS decrease over time means that the treatment is effective in decreasing GC toxicity level, compared to placebo which may show fluctuation of CIS over time. Negative score reflects that toxicities present at baseline (or occurring during the trial) resolved over the treatment period.

The steps to calculate the CWS and AIS at Week 24 and Week 52 are described below.

**Step 1:** Calculate domain-specific worsening score (for computing CWS in Step 2) and improvement score (for computing AIS in Step 2) at each visit.

For Domains without sub-items (Body Weight, Glucose Metabolism, Blood Pressure, Lipid Metabolism, Bone Health and Steroid Myopathy),

- a) For worsening score, only consider positive domain-specific score at each visit. For domain with a negative domain-specific score, the worsening score will be 0.
- b) For improvement score, all domain-specific scores (could be positive or negative) at each visit will be considered.

The Skin and Neuropsychiatric domains both have sub-items. For the Skin domain, these are Acneiform Rash, Easy Bruising, Hirsutism, Atrophy/Striae, and Erosions/tears/ulcerations. For the Neuropsychiatric domain, these are Insomnia, Depression, Mania, and Cognitive Impairment.

- a) For worsening score, only the item with the highest weight is scored for any GTI interval (typically three months) with the CWS. As an example, if neither insomnia nor depression were present at the baseline visit but there is now mild Insomnia and moderate depression present at follow-up, then only the moderate depression is scored (+63 points).
- b) For improvement score, improvement as well as worsening can be recorded. Because it is conceivable that one item might improve while another worsens, the item of greatest improvement (highest absolute weight) and the item of greatest worsening (highest weight) are recorded for given GTI interval.

For Infection Domain, the worsening score and improvement score handle the scoring of infections differently, because the CWS and AIS reflect reciprocal measures of GC toxicity.

- a) For worsening score, the most severe infection in every GTI interval is scored.
- b) For improvement score, only the most severe infection occurring over the course of the entire trial is scored.

**Step 2:** Calculate composite worsening score and improvement score at each visit\_by summing the 9 domain-specific score.

a) For composite worsening score, sum the 9 domain-specific worsening scores.

b) For composite improvement score, sum the 9 domain-specific improvement scores.

**Step 3:** Calculate cumulative GTI scores by summing composite scores across visits.

- a) For CWS at Week 24, summing composite GTI worsening score at Week 12 and Week 24.
- b) For CWS at Week 52, summing composite GTI worsening score at Week 12, Week 24, Week 40, and Week 52.
- c) For AIS at Week 24, summing composite GTI improvement score at Week 12 and Week 24.
- d) For AIS at Week 52, summing composite GTI improvement score at Week 12, Week 24, Week 40, and Week 52.

Table 4 – The Glucocorticoid Toxicity Index

| Composite GTI | ltem<br>weight | Specific List <sup>1</sup> |
|---|---|---|
| 1.BMI | | |
| Decrease by >/= 5 BMI units | -36 | Major increase in BMI |
| Decrease by >2 but <5 BMI units | -21 | |
| No significant change (+/- 2 BMI units) | 0 | |
| Increase of >2 to <5 BMI units | 21 | |
| Increase of 5 or more BMI units | 36 | |
| 2.Glucose tolerance | | |
| Improvement in HbA1c AND decrease in medication | -44 | Diabetic retinopathy |
| Improvement in HbA1c OR decrease in medication | -32 | Diabetic nephropathy |
| No significant change | 0 | Diabetic neuropathy |
| Increase in HbA1c OR increase in medication | 32 | |
| Increase in HbA1c AND increase in medication | 44 | |
| 3.Blood pressure | | |
| Improvement in BP AND decrease in medication | -44 | Hypertensive emergency |
| Improvement in BP OR decrease in medication | -19 | Posterior reversible encephalopathy |
| No significant change | 0 | syndrome |
| Increase in BP OR increase in medication | 19 | |
| Increase in BP AND increase in medication | 44 | |
| 4.Hyperlipidemia | | |
| Decrease in LDL AND decrease in medication | -30 | |
| Decrease in LDL OR decrease in medication | -10 | |
| No significant change | 0 | |
| Increase in LDL OR increase in medication | 10 | |
| Increase in LDL AND increase in medication | 30 | |
| 5.Bone Health (BMD) | | |
| Increase in BMD (gain of more than 3%) | -29 | Major decrease in bone density |
| No significant change in BMD (+/- 3%) | 0 | Insufficiency fracture |

| Composite GTI | ltem<br>weight | Specific List <sup>1</sup> |
|---|---|---|
| Decrease in BMD (loss of more than 3%) | 29 | |
| 6.Steroid myopathy | | |
| Moderate weakness to none | -63 | Severe steroid myopathy |
| Moderate to Mild weakness | -54 | |
| Mild weakness to none | -9 | |
| No significant change | 0 | |
| None to Mild weakness (without functional limitation) | 9 | |
| Mild to Moderate weakness | 54 | |
| None to Moderate weakness (with functional limitation) | 63 | |
| 7.Skin steroid-related Toxicity | | |
| Decrease in Skin Toxicity - Moderate to None | -26 | Severe skin toxicity |
| Decrease in Skin Toxicity - Moderate to Mild | -18 | |
| Decrease in Skin Toxicity - Mild to None | -8 | |
| No significant change | 0 | |
| Increase in Skin Toxicity - None to Mild | 8 | |
| Increase in Skin Toxicity - Mild to Moderate | 18 | |
| Increase in Skin Toxicity - None to Moderate | 26 | |
| 8.Neuropsychiatric - steroid related symptoms | | |
| Decrease in NP Toxicity - Moderate to None | -74 | Psychosis |
| Decrease in NP Toxicity - Moderate to Mild | -63 | GC-induced violence |
| Decrease in NP Toxicity - Mild to None | -11 | Other severe neuropsychiatric |
| No significant change | 0 | symptoms |
| Increase in NP Toxicity - None to Mild | 11 | |
| Increase in NP Toxicity - Mild to Moderate | 63 | |
| Increase in NP Toxicity - None to Moderate | 74 | |
| 9.Infection | | |
| No infection | 0 | Grade IV infection |
| Oral or vaginal candidiasis or non-complicated zoster ( <grade3)< td=""><td>19</td><td>Grade V infection</td></grade3)<> | 19 | Grade V infection |
| Grade 3, 4, or 5 infection | 93 | |

<sup>&</sup>lt;sup>1</sup> Maximum weight is given for specific list events in Blood pressure, Steroid myopathy, Skin toxicity, Neuropsychiatric and Infection domains at each visit. For the rest of domains, specific list events will not affect the corresponding domain specific score.

# 2.1.4 Safety endpoints

The safety analysis will be based on the reported adverse events (AEs), serious AEs (SAEs) and adverse events of special interest (AESIs) including but not limited to neutropenia, thrombocytopenia, elevations in hepatic enzymes leading to permanent discontinuation and

tuberculosis, and other opportunistic infections. Other safety information, such as clinical laboratory data and vital signs will also be assessed.

#### Observation period

The observation period will be divided into 4 epochs:

- The **screening** epoch is defined as the time from the signed informed consent date up to the time prior to first dose of SC IMP.
- The **treatment** epoch is defined as the time from the first dose of the IMP to the last dose of the SC IMP in the DB period +13 days.
- The **residual treatment** epoch is defined as the time from the end of TREATMENT epoch to the last dose of the SC IMP +60 days.

The **post-treatment** epoch is defined as the time after the last dose of SC IMP +60 days. The rationale of having "last dose of SC IMP +60 days" as the end of follow-up epoch is to capture the events observed within an approximately 5 half-lives of the last sarilumab SC IMP.

The treatment-emergent adverse event (TEAE) period includes both **treatment** and **residual treatment** epochs.

#### 2.1.4.1 Adverse events variables

## Adverse event observation period

- Pre-treatment AEs are AEs that developed or worsened or became serious from the signed informed consent date up to first administration of SC IMP
- TEAEs are AEs that developed or worsened or became serious during the TEAE period
- Post-treatment AEs are AEs that developed or worsened or became serious during the post-treatment period

All AEs (including SAEs and AESIs) will be coded to a "LLT", "PT", "HLT", "HLGT", and associated primary "SOC" using the version of MedDRA currently in effect at Sanofi at the time of database lock.

The occurrence of AEs (including SAEs and AESIs) will be recorded from the time of signed informed consent until the end of the study.

Any SAE brought to the attention of the Investigator at any time after the end of the study for the patient and considered by him/her to be caused by the IMP with a reasonable possibility, should be reported to the monitoring team.

# Adverse event of special interest (AESI)

Adverse events of special interest will be flagged in the database. The AESIs and its search criteria are listed in Table 5 below:

08-Jan-2021 Version number: 1

Table 5 - Protocol defined AESIs and search criteria

| AESI flag | Search criteria |
|---|---|
| Clinically significant infections including: | Reported by the investigators on the AE CRF page with AESI box ticked. |
| ANC decrease leading to permanent discontinuation Thrombocytopenia leading to permanent discontinuation ALT >= 3xULN | |
| Pregnancy | CRF checkbox: Pregnancy |
| Overdose | CRF checkbox: Symptomatic Overdose |

#### 2.1.4.2 Deaths

The deaths per the observation period will be summarized.

- Death on-treatment: deaths occurring during the treatment period (i.e., treatment Epoch)
- Death during follow-up: deaths occurring during the residual treatment period
- Death post-treatment: deaths occurring during the post-treatment period

## 2.1.4.3 Laboratory safety variables

Clinical laboratory data will include hematology, clinical chemistry, and urinalysis. Clinical laboratory values will be converted to standard international units; international units will be used in all listings and tables. In addition, the lipids parameters will also be summarized in US units.

Hematology and chemistry data will be collected at screening, baseline, Weeks 4,12, 24, 40, and 52, and/or early termination unless otherwise specified. The laboratory parameters will be classified as follows:

- Hematology
  - Red blood cells and platelets and coagulation: hemoglobin, hematocrit, platelet count, red blood cell (RBC) count, and RBC morphology (if RBC count is abnormal).
  - White blood cells: white blood cell (WBC) count and WBC differential (neutrophils, lymphocytes, monocytes, basophils, eosinophils).
- Clinical chemistry
  - **Metabolism:** fasting lipids (total cholesterol, high density lipoprotein cholesterol (HDL-C), low density lipoprotein cholesterol (LDL-C), ratio of HDL-C versus LDL-C (HDL-C:LDL-C), triglycerides), total proteins, CRP, fasting glucose, and hemoglobin A1c (HbA1c).

- Electrolytes: sodium, potassium, chloride, calcium, phosphate, and bicarbonate.
- **Renal function:** creatinine, creatinine clearance, uric acid, and blood urea nitrogen (BUN).
- **Liver function:** alanine aminotransferase (ALT)/SGPT, aspartate aminotransferase (AST)/SGOT, alkaline phosphatase (ALP), albumin, total bilirubin, conjugated and unconjugated bilirubin, and lactate dehydrogenase (LDH).
- **Pregnancy test:** Serum β-hCG for all women of childbearing potential (screening only).
- **TB screen:** QuantiFERON®-TB Gold evaluation.
- **Hepatitis screen:** Hepatitis B and C serology, human immunodeficiency virus serology.

Urine samples will be collected as follows:

• Urinalysis - dipstick: pH, specific gravity, blood, glucose, protein, nitrates, leukocyte esterase, and bilirubin. If any parameter on the dipstick is abnormal, a urine sample was to be sent to the central laboratory for testing.

A urine pregnancy test was done for all women of childbearing potential at baseline, all visits up to Week 52 or early termination.

# 2.1.4.4 Vital signs variables

Vital signs variables include heart rate, systolic blood pressure, and diastolic blood pressure, height, weight, and body temperature.

#### 2.1.4.5 Antinuclear antibodies

Antinuclear antibodies (ANA) will be measured at baseline and EOT visits.

# 2.1.5 Immunogenicity endpoints

The immunogenicity blood samples will be collected before injection during the same visit according to the Study Flow Chart (Appendix A).

Samples analyzed in the antidrug antibody (ADA) assay will be categorized as either positive or negative, and in the case of a positive result will be further characterized as either neutralizing or non-neutralizing.

<u>ADA positive patient</u> is defined as patient with at least one treatment-emergent or treatment-boosted ADA positive sample during the TEAE period, where

- Treatment-emergent ADA positive patient is defined as a patient with non-positive assay (meaning negative or missing) response at baseline but with a positive assay response during the TEAE period.
- Treatment-boosted ADA positive patient is defined as a patient with a positive ADA assay response at baseline and with at least a 4-fold increase in titer compared to baseline during the TEAE period.

<u>ADA negative patient</u> is defined as patient without a treatment-emergent or treatment-boosted ADA positive sample during the TEAE period.

A treatment-emergent positive response is further classified as persistent or transient.

<u>Persistent ADA response:</u> treatment-emergent ADA detected at two or more consecutive sampling time points during the TEAE period, where the first and last ADA positive samples are separated by a period of at least 16 weeks. Also persistent in case last sample analyzed is positive.

<u>Transient ADA response:</u> A treatment-emergent response that is not determined to be persistent.

#### 2.1.6 Pharmacokinetic variables

The blood samples for the determination of functional sarilumab concentrations in serum will be collected before injection during the same visit according to the Study Flow Chart (refer to Section 1.2 in the study protocol) and at or near the onset and completion of the occurrence of a SAE.

## 2.1.7 Pharmacodynamic/genomics endpoints

Blood samples (DNA and genetic RNA) will be collected from each consenting patient to participate in the pharmacogenomics substudy. Details of any analysis will be described in a separate plan.

## 2.1.8 Other efficacy endpoints

Quality-of-life endpoints

Other efficacy endpoints in the clinical outcome assessments will be summarized. Patients are asked to complete the following patient-reported outcome (PRO) questionnaires described below at Visit 2 (baseline visit), Visit 6 (Week 12), Visit 9 (Week 24), and Visit 12 (Week 52).

## **Patient-Reported Outcomes**

## Short Form 36 Version 2 (SF-36 V2)

The SF-36 V2 is a multi-purpose, short-form health survey with 36 questions. It yields scores for eight domains (Physical Functioning, Role-Physical, Bodily pain, General health, Vitality, Social Functioning, Role-Emotional, and Mental Health, each scale is scored from 0 to 100 where higher scores indicate better health and well-being), as well as two summary measures of physical and mental health: the Physical Component Summary (PCS) and Mental Component Summary (MCS).

The scoring process is summarized below:

- Enter item response data.
- Recode item response values.
- Determine health domain scale raw scores.
- Transform health domain scale raw scores to 0 to 100 scores.
- Transform health domain scale 0 to 100 to normal-based scores.
- Score physical and mental component summary measures.

The following table shows the construction and summary measures of the SF-36 scales:

Table 6 - SF-36 V2 measurement model

| Summary measures | Scales | Items |
|---|---|---|
| Physical Component | Physical Functioning (PF) | 3a, 3b, 3c, 3d, 3e, 3f, 3g, 3h, 3i, 3j |
| Summary (PCS)* | Role-Physical (RP) | 4a, 4b, 4c, 4d |
| | Bodily Pain (BP) | 7, 8 |
| | General Health (GH) | 1, 11a, 11b, 11c, 11d |
| Mental Component | Vitality (VT) | 9a, 9e, 9g, 9i |
| Summary (MCS)* | Social Functioning (SF) | 6, 10 |
| | Role-Emotional (RE) | 5a, 5b, 5c |
| | Mental Health (MH) | 9b, 9c, 9d, 9f, 9h |

<sup>\*</sup>MCS and PCS derived from the eight scales

The score of each of the 36 items is collected in CRF. Appendix G provides the SAS code to calculate the eight scales, the two summary measure scores and the standardized summary scores.

The PCS and MCS summary measure scores will be computed if at least 50% of the component scales are available. The scale scores will be computed if at least 50% of items are available within the corresponding scale. The missing items will be imputed by the mean of available items.

Change from baseline in SF-36 scores (physical component summary score and mental component summary score as well as the eight domains) at each visit will be analyzed.

# Functional Assessment of Chronic Illness Therapy Fatigue (FACIT-Fatigue)

The FACIT-Fatigue will be used to assess fatigue. The FACIT-Fatigue is a 13-item questionnaire rated 0 to 4 originally developed to measure fatigue in patients with cancer and is widely used in rheumatoid arthritis patients to demonstrate good consistency and sensitivity to change. The patient will be asked to answer 13 questions rated 0 to 4 (0 = not at all, 1 = a little bit, 2 = somewhat, 3 = quite a bit, 4 = very much). The fatigue scale has 13 items, with 52 as the highest possible score. A higher score in the fatigue scale corresponds to a lower level of fatigue and indicates better Quality of Life.

To calculate the FACIT-fatigue score, the response scores on negatively phrased questions are reversed and then the 13 item responses are added. Eleven items with responses have their scores reversed (item score = 4 – response, if the response is not missing), and two items (items 7 and 8) have their responses unchanged (Appendix E). All items are added so that higher scores correspond to less fatigue. In cases where individual questions are skipped, scores are prorated using the average of other answers in the scale.

FACIT-Fatigue = 13 \* [sum (reversed items) + sum (items 7 and 8)] / number of answered items

## EuroQol 5 Dimension 3 Level (EQ-5D-3L)

The EQ-5D-3L is a standardized, generic measure of health outcome (3). EQ-5D is designed for selfcompletion by patients. Instructions to respondents are included in the questionnaire. The EQ5D is specifically included to address concerns regarding the health economic impact of RA, which have been considered in cost effectiveness arguments. The EQ-5D-3L comprises five questions on mobility, self-care, pain, usual activities, and psychological status with three possible answers for each item (1 = no problem, 2 = moderate problems, 3 = severe problems) and a vertical visual analog scale that allows the patients to indicate their health state today that can range from 0 (worst imaginable) to 100 (best imaginable).

The 5 dimensional 3-level systems are converted into a single index utility score. Values for the 243 theoretically possible health states defined by the EuroQol classification are calculated using a regression model and weighted according to the social preferences of the GB population. The minimum value for the single index utility score is -0.594, which corresponds to a level 3 (severe problems) for mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The maximum value for this index is 1.0, which corresponds to a full health (level 1 [no problem] for mobility, self-care, usual activities, pain/discomfort and anxiety/depression).

The VAS records the respondent's self-rated health on a vertical visual analogue scale. The VAS "thermometer" has endpoints of 100 (Best imaginable health state) at the top and 0 (Worst imaginable health state) at the bottom. This information can be used as a quantitative measure of health outcomes as judged by the individual respondents. EQ 5D self-reported VAS data generates information on the self-perceived overall health-related quality of life.

Appendix F provides the SAS code to derive the index utility score using GB based population.

# Health Assessment Questionnaire Disease Index (HAQ-DI)

## • Patient's Assessment of Physical function

The HAQ-DI is a standardized questionnaire developed to assess physical functional status in adults with arthritis but is now commonly used among many rheumatologic conditions. The HAQ-DI, with the past week as the time frame, focuses on whether the respondent "is able to…" do the activity and covers eight categories in 20 items: dressing and grooming, arising, eating, walking, hygiene, reach, grip and activities, for which there are at least two questions by category. The four responses for the HAQ-DI questions are graded as follows: without any difficulty=0; with some difficulty=1; with much difficulty=2; and unable to do=3. To calculate the Standard HAQ-DI Score (With Aids/Devices), there are 3 steps:

- 1. Sum the eight category scores by using the highest sub-category score from each category.
- For example, in the category EATING there are three sub-category items. A patient responds with a 1, 2, and 0, respectively; the category score is 2.
- 2. Adjust for use of aids/devices and/or help from another person when indicated.
- When there are NO aids or devices or help indicated for a category, the category's score is not modified.
- When aids or devices or help ARE indicated by the patient:
  - Adjust the score for a category by increasing a 0 or a 1 to a 2.
  - If a patient's highest score for that sub-category is a 2 it remains a 2, and if a 3, it remains a 3.
  - The data entered at field "Other specify" will not be used for score adjustment.
- 3. Divide the summed category scores by the number of categories answered (must be a minimum of 6) to obtain a HAQ-DI score of 0 to 3 (3=worst functioning).

A HAQ-DI score cannot be calculated validly when there are scores for less than six of the eight categories. If there are less than 6 categories completed, a HAQ-DI cannot be computed, whether the missing categories are due to missing values or they do not apply to the respondent. HAQ-DI disability index scoring ranges between 0 and 3 with higher score indicating greater disability. A high HAQ-DI score has been found to be a strong predictor of morbidity and mortality in RA. A 0.22 unit difference is considered clinically meaningful.

In addition to the above, the HAQ-DI has two additional questions to measure pain and global assessment described below.

## • Patient's Assessment of Pain

Patients will be requested to indicate their pain intensity due to PMR using a 100 mm horizontal VAS to the question "How much pain have you had IN THE PAST WEEK?", where 0 is considered "No pain" and 100 "the worst pain you can imagine".

To obtain the patient score, using a metric ruler, measure the distance in centimeters from the left anchor (at base zero) to their mark and multiply by 0.2. This converts the number of centimeters into the appropriate score and yields a score from 0 to 3. For example, the mark is at 8 centimeters  $-8 \times 0.2 = a$  pain score of 1.6.

In case a 0-100 mm scale is used, pain severity coding translations follow below:

## PAIN SEVERITY CODING TRANSLATIONS

| Measurement (m) = Score | Measurement (m) = Score [continue] |
|-------------------------|------------------------------------|
| 0 = 0 | 7.8 - 8.2 = 1.6 |
| 0.1 - 0 .7 = 0.1 | 8.3 - 8.7 = 1.7 |
| 0.8 - 1.2 = 0.2 | 8.8 - 9.2 = 1.8 |
| 1.3 - 1.7 = 0.3 | 9.3 - 9.7 = 1.9 |
| 1.8 - 2.2 = 0.4 | 9.8 - 10.2 = 2.0 |
| 2.3 - 2.7 = 0.5 | 10.3 - 10.7 = 2.1 |
| 2.8 - 3.2 = 0.6 | 10.8 - 11.2 = 2.2 |
| 3.3 - 3.7 = 0.7 | 11.3 - 11.7 = 2.3 |
| 3.8 - 4.2 = 0 .8 | 11.8 - 12.2 = 2.4 |
| 4.3 - 4.7 = 0 .9 | 12.3 - 12.7 = 2.5 |
| 4.8 - 5.2 = 1.0 | 12.8 - 13.2 = 2.6 |
| 5.3 - 5.7 = 1.1 | 13.3 - 13.7 = 2.7 |
| 5.8 - 6.2 = 1.2 | 13.8 - 14.2 = 2.8 |
| 6.3 - 6.7 = 1.3 | 14.3 - 14.7 = 2.9 |
| 6.8 - 7.2 = 1.4 | 14.8 - 15.0 = 3.0 |

## • Patient's Global Assessments of Disease Activity

Patient's global assessments of their current disease activity will be rated on an anchored 100 mm horizontal VAS, with the given instruction to "Please rate how well you are doing on a scale of 0 to 100 (0 represents "very well" and 100 represents "very poor" health)".

It is scored similarly to the VAS Pain Scale.

# **Clinician-Reported Outcomes**

## Physician's Global Assessments of Disease Activity - Visual Analog Scale [MD-VAS]

Physician's global assessments of the patient's current disease activity will be assessed on an anchored 100 mm horizontal VAS where 0 is considered the best disease activity (no disease activity) and 100 the worst (most disease activity).

#### 2.2 DISPOSITION OF PATIENTS

This section describes patient disposition for both patient status and the patient populations.

Screened patients are defined as all patients who signed the informed consent.

Randomized patients consist of all patients who signed informed consent with a treatment kit number allocated and recorded in the Interactive Voice Response System/Interactive Web Response System database, regardless of whether the treatment kit was used or not.

For patient status in the DB treatment period, the total number of patients for each one of the following categories will be presented in the clinical study report (CSR) using a summary table:

- Screened patients
- Screen failure patients and reasons for screen failure
- Non-randomized but treated patients
- Randomized patients
- Randomized but not treated patients
- Randomized and treated patients
- Patients who completed SC IMP treatment up to Week 24
- Patients who discontinued SC IMP treatment before Week 24 and the reasons for permanent treatment discontinuation
- Patients who completed 52-week SC IMP study treatment period
- Patients who discontinued from 52-week study treatment period and the reasons for permanent SC IMP treatment discontinuation
- Patients who completed the study
- Patients who discontinued the study and the reasons for study discontinuation
- Patients who took CS rescue therapy
- Subject status at end of study visit

For all categories of patients (except for the screened and non-randomized categories) percentages will be calculated using the number of randomized patients as the denominator. Reasons for discontinuation with regards to SC IMP treatment will be presented in tables giving numbers and percentages by treatment group.

A patient is considered as lost to follow-up at the end of the study if he/she is not assessed at the end of study visit.

All critical or major deviations potentially impacting efficacy analyses, randomization and drug dispensing irregularities and other major/critical deviations will be summarized in tables giving numbers and percentages of deviations by treatment groups.

Additionally, the analysis populations for safety, efficacy, PK, and immunogenicity will be summarized in a table by patient counts based on the randomized populations (See definitions in Section 2.3).

• Efficacy population

- Safety population
- PK population

OR

ADA population

# 2.2.1 Randomization and drug dispensing irregularities

Randomization and drug-dispensing irregularities occur whenever:

1. A randomization is not in accordance with the protocol-defined randomization method, such as a) an ineligible patient is randomized, b) a patient is randomized based on an incorrect stratum, c) a patient is randomized twice, or d) in a dynamic randomization scheme the treatment assignment is, in fact, not random, due to a computer program error.

2. A patient is dispensed an IMP kit not allocated by the protocol-defined randomization, such as a) a patient at any time in the study is dispensed a different treatment kit than as randomized (which may or may not contain the correct-as-randomized IMP), or b) a nonrandomized patient is treated with IMP reserved for randomized patients.

Randomization and drug-dispensing irregularities will be monitored throughout the study and reviewed on an ongoing basis.

All randomization and drug-dispensing irregularities will be documented in the CSR. If the number of irregularities is large enough to make a tabular summary useful, the irregularities will be categorized and summarized among randomized patients (number and percentages). Nonrandomized, treated patients will be described separately.

Randomization and drug-dispensing irregularities to be prospectively identified include but are not limited to:

Table 7 - Randomization and Drug Allocation Irregularities

# Randomization and Drug Allocation Irregularities

Kit dispensation without IVRS transaction Erroneous kit dispensation Kit not available Randomization by error Subject randomized twice Forced randomization Subject switched to another site

IVRS=Interactive Voice Response System

#### 2.3 ANALYSIS POPULATIONS

The randomized population includes any patient who has been allocated to a randomized treatment regardless of whether the treatment kit was used.

Patients treated without being randomized will not be considered randomized and will not be included in any efficacy population.

For any patient randomized more than once, only the data associated with the first randomization will be used in any analysis population. The safety experience associated with any later randomization will be assessed separately.

The safety experience of patients treated and not randomized will be reported separately, and these patients will not be in the safety population.

# 2.3.1 Efficacy populations

Week 52 Analysis set: The primary endpoint for the study is sustained remission at Week 52. Based on patients' enrollment dates and the study discontinuation plan, not all the patients had an opportunity to complete the 52-week treatment period. For the cohort of patients who did not have an opportunity to complete the 52-week treatment period, it is not meaningful to define the endpoint of sustained remission at Week 52. Therefore, the analysis of primary endpoint will be limited to the Week 52 Analysis set, which includes the cohort of patients who had an opportunity to complete the 52-week treatment period. This cohort of patients is defined as the patients with a randomization date prior to *Oct 16*, *2019* (i.e., *Oct 13*, *2019*+3 days IMP administration time window, where *Oct 13*, *2019* is 1-year before the targeted last patient last EOT visit date [i.e., *Oct 13*, *2020*] according to the study discontinuation plan), which contains a total of 36 patients (out of 83 randomized patients).

For the same reason, the analysis of secondary endpoint of cumulative GTI scores at Week 52 will also be limited to the cohort of patients who had an opportunity to complete the 52-week treatment period.

For the rest of the efficacy endpoints, the primary analysis population will be the ITT population as defined in Section 2.3.1.1.

#### 2.3.1.1 Intent-to-treat population

The intent-to-treat (ITT) population is the randomized population analyzed according to the treatment group allocated by randomization.

#### 2.3.2 Safety population

The safety population is defined as randomized population who actually received at least 1 dose or part of a dose of the SC IMP, analyzed according to the treatment actually received

#### In addition:

- Nonrandomized but treated patients will not be part of the safety population; however, their safety data will be presented separately
- Randomized patients for whom it is unclear whether they took the IMP will be included in the safety population as randomized

• For patients receiving more than one SC IMP during the trial, the treatment group allocation for as-treated analysis will be the treatment group for which the patient received the majority of doses. In such cases, individual patient listings will be provided for each treatment group with treatment start and end date for each treatment exposed.

#### 2.3.3 Pharmacokinetics and ADA populations

The PK population will consist of all patients in the safety population with at least one post-dose, non-missing serum sarilumab concentration value. The ADA population will consist of all patients in the safety population with at least one post-dose, evaluable ADA sample. Patients will be analyzed according to the treatment actually received.

#### 2.4 STATISTICAL METHODS

## 2.4.1 Demographics and baseline characteristics

Continuous data will be summarized using the number of available data, mean, standard deviation (SD), median, minimum, and maximum for each treatment group. Categorical and ordinal data will be summarized using the number and percentage of patients in each treatment group.

Parameters will be summarized based on the randomized populations.

Parameters described in Section 2.1.1 will be summarized by treatment group and overall using descriptive statistics.

Medical and surgical history will be summarized by SOC and PT sorted by internationally agreed order of SOC and by the decreasing frequency of PT within SOC in total group (including all the randomized patients). P-values on demographic and baseline characteristic data will not be calculated.

No specific description of the safety parameters will be provided at baseline. If relevant, the baseline values will be described along with each safety analysis.

#### 2.4.2 Prior or concomitant medications

The prior and concomitant medications will be summarized based on the randomized populations as follows:

- Prior medications discontinued before the first dose of IMP in the DB period
- Prior medications that continued at the time of the first dose of IMP in the DB period
- Concomitant medications

Medications will be summarized by treatment group according to the WHO-DD dictionary, considering the first digit of the anatomic category (ATC) class (anatomic category) and the
generic names. All ATC codes corresponding to a medication will be summarized. Patients will be counted once in each ATC category (anatomic or therapeutic) linked to the medication; therefore, patients may be counted several times for the same medication.

In addition, the following summaries will also be provided:

- Vaccines (prior and concomitant vaccines will be summarized separately)
- Other prior DMARDs/immunosuppressive agents taken since diagnosis of GCA and discontinued before the first dose of IMP

The table for prior medications will be sorted by decreasing frequency of anatomic category followed by all other generic names based on the overall incidence across treatment groups. In case of equal frequency regarding anatomic categories (respectively, generic names), alphabetical order will be used.

The tables for concomitant medications will be sorted by decreasing frequency of anatomic category followed by all other generic names based on the incidence of the total group (including all the randomized patients). In case of equal frequency regarding anatomic categories (respectively, generic names), alphabetical order will be used.

# 2.4.3 Extent of investigational medicinal product exposure and compliance

The extent of SC IMP exposure and compliance will be assessed and summarized by actual treatment group within the safety population (Section 2.3.2).

# 2.4.3.1 Extent of investigational medicinal product exposure

The extent of SC IMP exposure will be assessed by the duration of SC IMP exposure and actual dose information.

The duration of SC IMP exposure is defined as last DB dose date – first DB dose date +14 days, regardless of unplanned intermittent discontinuations (see Section 2.5.3 for calculation in case of missing or incomplete data).

Duration of SC IMP exposure will be summarized descriptively as a quantitative variable (number, mean, SD, median, minimum, and maximum). In addition, duration of treatment exposure will also be summarized categorically by numbers and percentages for each of the following categories and cumulatively according to these categories:  $\le 4$  weeks, >4 and  $\le 8$  weeks, >8 and  $\le 12$  weeks, >12 and  $\le 16$  weeks, >16 and  $\le 20$  weeks, >20 and  $\le 24$  weeks, >24 and  $\le 32$  weeks, >32 and  $\le 40$  weeks, >40 and  $\le 52$  weeks and >52 weeks.

Additionally, the cumulative duration of treatment exposure, defined as the sum of patients' duration of treatment exposure and expressed in patient years, will be provided.

#### 2.4.3.2 Compliance

A given administration will be considered noncompliant if the patient did not take the planned dose of treatment as required by the protocol. No imputation will be made for patients with missing or incomplete data.

Percentage of compliance for SC IMP will be defined as the number of administrations the patient was compliant divided by the total number of administrations the patient was planned to take on or before the last dose date during the DB treatment period.

Percentage of compliance for oral IMP compliance rate will be defined as the total number of days patient with partial or complete oral IMP intake divided by total number of days between the first oral IMP intake date and day prior to rescue therapy start date or EOT date which is earlier.

Treatment compliance percentages will be summarized descriptively as quantitative variables (number, mean, SD, median, minimum, and maximum). The percentage of patients whose compliance is <80% will be summarized.

Cases of overdose (administering two or more doses of sarilumab or its matching placebo in less than 11 calendar days) will constitute AESI and will be listed as such. More generally, dosing irregularities will be listed in Section 2.2.1.

#### 2.4.4 Analyses of efficacy endpoints

The analyses of efficacy endpoints will be descriptive in nature. For majority of the efficacy endpoints, only descriptive summary statistics will be provided by 4 treatment groups. For the primary and some selected important secondary endpoints, summary statistics and formal statistical tests on between group comparisons (with 95% CI and p-value) will be provided for the 2 combined treatment groups (ie, 2 sarilumab groups combined versus 2 placebo groups combined); no formal comparisons will be performed between 4 individual treatment groups due to the small sample size.

# 2.4.4.1 Analysis of primary and additional efficacy endpoint(s)

The analysis of primary endpoint of sustained remission at Week 52 will be limited to the cohort of patients who had an opportunity to complete the 52-week treatment period (i.e., Week 52 Analysis set).

The proportion of patients achieving sustained remission at Week 52 will be summarized using counts and percentages by the 4 treatment groups. In addition, the treatment effects between the combined sarilumab (group A+B) group and the combined placebo group (Group C+D) will be compared using a Cochran-Mantel-Haenszel (CMH) test stratified by prednisone dose at baseline (<30 mg/day or ≥30 mg/day).

The additional endpoint of sustained remission at Week 24 will be analyzed in the same fashion in the ITT population.

# Sensitivity analysis excluding acute phase reactants:

Sensitivity analysis will be performed for the primary endpoint by removing the acute phase reactants (CRP and ESR) from the definition to mitigate against the possibility of biasing the results due to the known PD effect of sarilumab on acute phase reactants.

Patients achieving sustained remission at Week 52 (or Week 24) excluding acute phase reactants is defined by having met all of the following parameters:

- Achievement of disease remission not later than Week 12. Disease remission is defined as resolution of signs and symptoms of GCA.
  - **AND**
- Absence of disease flare from Week 12 through Week 52 (or Week 24). **Flare** is defined as recurrence of signs and symptoms attributable to active GCA plus an increase in CS dose due to GCA.

**AND** 

• Successful adherence to the prednisone taper from Week 12 through Week 52 (or Week 24).

The sensitivity analysis will be performed in the same fashion as for the primary endpoint. Descriptive statistics (i.e., counts and percentages) will be provided for the three individual components.

#### **Subgroup analyses:**

No subgroup analyses will be performed due to the small sample size.

# 2.4.4.2 Analyses of secondary efficacy endpoints

# Components of sustained remission composite measure at Week 52 and Week 24

Descriptive statistics (i.e., counts and percentages) will be provided for the following binary variables by treatment groups:

- Patients who achieve disease remission by Week 12
- Patients who have absence of disease flare from Week 12 through Week 52 (or Week 24)
- Patients who have normalization of CRP (decrease to <10 mg/L) with sustained normalization from Week 12 through Week 52 (or Week 24)
- Patients who successfully adhere to the prednisone taper from Week 12 through Week 52 (or Week 24)

# Total cumulative corticosteroid (including prednisone) dose

Descriptive statistics including the number of subjects, mean, and median of the total cumulative prednisone (or equivalent) dose will be presented for each treatment group. The difference between the medians and the corresponding 95% non-parametric confidence interval along with

p-value from the non-parametric Wilcoxon rank-sum test between the two combined treatment groups will also be provided.

The total cumulative CS dose will be based on the total number of days with complete or partial intake, no imputation will be done on missed tablets. Patients who received increased prednisone or equivalent in rescue therapy will be included in their original treatment groups.

In the scenario that a patient has already taken external CS for the disease before randomization on the day of randomization, the CS dose taken will be considered as the first dose of oral IMP. The first dose of prednisone per tapering regimen will be skipped, and the patient will take the second dose of prednisone on the next day.

#### Time to first GCA flare during the treatment period

Time (from randomization) to the first GCA flare after clinical remission up to Week 52 will be analyzed by Kaplan-Meier method providing the median, 25<sup>th</sup> and 75<sup>th</sup> percentiles (where possible) along with the 95% CI for the median. The comparison between the two combined groups will be performed using Cox proportional hazards model with prednisone dose at baseline (<30 mg/day or ≥30 mg/day) included as a covariate. Hazard ratio and the corresponding 95% CI and p-value will be provided.

### Composite GTI and Specific List

#### GTI analyses

Descriptive statistics including number, mean, SD, SE, median, minimum, and maximum will be provided by treatment group and by visit for domain-specific GTI score, composite GTI total score, composite worsening score and composite improvement score. For CWS and AIS at Week 52 and Week 24, analysis of covariance (ANCOVA) model with treatment (combined sarilumab groups and combined placebo groups), baseline glucocorticoid toxicity score and baseline prednisone dose (<30 mg/day or ≥30 mg/day) as fixed effects, will be used to test the difference of the least-square means (LS means) between the two combined groups. Difference in LS means and the corresponding 95% CI along with the p-value will be provided.

In addition, descriptive statistics (i.e., counts and percentages) will be provided for not worsening (CWS > 0), worsening (CWS  $\leq$  0), improved (AIS  $\leq$  0) and not improved (AIS  $\geq$ 0) at Week 52 and Week 24. Odds ratios and exact 95% CIs of not worsening versus worsening and improved versus not improved will be provided for the comparisons between the combined sarilumab groups and combined placebo groups as well.

Please note, the analysis of cumulative GTI scores (i.e., CWS and AIS) at Week 52 will be limited to the cohort of patients who had an opportunity to complete the 52-week treatment period (i.e., Week 52 Analysis set).

#### Analyses of items in Specific list

Number and percentage of patients with each item in specific list will be summarized by treatment groups and by visit.

# 2.4.4.3 Multiplicity issues

No adjustments for multiplicity will be applied for this study due to the small sample size and the fact that many patients will not have the opportunity to complete the planned 52-week treatment period. All reported p-values will be nominal.

# 2.4.5 Analyses of safety data

The summary of safety results will be presented by treatment groups.

#### General common rules

All safety analyses will be performed on the safety population as defined in Section 2.3.2, unless otherwise specified, using the following common rules:

- Safety data in patients who do not belong to the safety population (eg, exposed but not randomized) will be listed separately
- The baseline value is defined as the last available value prior to the first dose of study medication.
- The potentially clinically significant abnormality (PCSA) values are defined as abnormal values considered medically important by the Sponsor according to predefined criteria/thresholds based on literature review and defined by the Sponsor for clinical laboratory tests, vital signs, and ECG (PCSA in BTD-009536 version 3, see Appendix B)
- PCSA criteria will determine which patients had at least 1 PCSA during the TEAE period, taking into account all evaluations performed during the TEAE period, including nonscheduled or repeated evaluations. The number of all such patients will be the numerator for the on-treatment PCSA percentage
- The treatment-emergent PCSA denominator by group for a given parameter will be based on the number of patients assessed for that given parameter in the treatment-emergent adverse event period by treatment group on the safety population.
- For quantitative safety parameters based on central laboratory/reading measurements, descriptive statistics will be used to summarize results and change from baseline values by visit and treatment group. Summaries will include the endpoint value. The endpoint value is commonly defined as the value collected at the same day/time of the last dose of investigational product. If this value is missing, this endpoint value will be the closest one prior to the last dose intake.
- Analyses of the safety variables will be essentially descriptive and no systematic testing is planned.

## 2.4.5.1 Analyses of adverse events

#### **Generalities**

The primary focus of AE reporting will be on TEAEs. Pre-treatment and post-treatment AEs will be described separately.

If an AE date/time of onset (occurrence, worsening, or becoming serious) is incomplete, an imputation algorithm will be used to classify the AE as pre-treatment, or TEAE, or post-treatment AE. The algorithm for imputing date/time of onset will be conservative and will classify an AE as treatment-emergent unless there is definitive information to determine it is pre-treatment or post-treatment. Details on classification of AEs with missing or partial onset dates are provided in Section 2.5.3.

Adverse event incidence tables will present by SOC, HLGT, HLT, and PT, sorted in SOC internationally agreed order and then alphabetical order, and present the number (n) and percentage (%) of patients experiencing an AE by treatment group. Multiple occurrences of the same event in the same patient will be counted only once in the tables within a treatment phase. The denominator for computation of percentages is the safety population within each treatment group.

The tables by primary SOC and PT will be sorted by internationally agreed order of SOC and decreasing frequency of PT within SOC. Sorting will be based on results for the sarilumab 200mg arm.

# Analysis of all treatment-emergent adverse events

The following TEAE summaries will be generated for the safety population.

- Overview of TEAEs, summarizing number (%) of patients with any
  - TEAE
  - Serious TEAE
  - TEAE leading to death
  - TEAE leading to permanent treatment discontinuation
- All TEAEs by primary SOC, HLGT, HLT, and PT, showing number (%) of patients with at least one TEAE sorted by SOC internationally agreed order. The other level (HLGT, HLT, PT) will be presented in an alphabetic order.
- All TEAEs by primary SOC and PT, showing number (%) of patients with at least one TEAE, sorted by SOC internationally agreed order and decreasing incidence of PTs within SOC. This sorting order will be applied to all other tables, unless otherwise specified.
- All TEAEs by primary SOC, showing number (%) of patients with at least one TEAE, sorted by internationally agreed order of primary SOC.

- All TEAEs by relationship, presented by primary SOC, HLGT, HLT, and PT, showing number (%) of patients with at least one TEAE, sorted by SOC internationally agreed order. The other level (HLGT, HLT, PT) will be presented in an alphabetic order.
- All TEAEs by maximal severity, presented by primary SOC and PT, showing number (%) of patients with at least one TEAE by severity (ie, mild, moderate, or severe), sorted by sorting order defined above.

### Analysis of all treatment emergent serious adverse event(s)

- All treatment-emergent SAEs by primary SOC, HLGT, HLT, and PT, showing number (%) of patients with at least one serious TEAE, sorted by SOC internationally agreed order. The other level (HLGT, HLT, PT) will be presented in an alphabetic order.
- All treatment-emergent SAEs by primary SOC and PT, showing number (%) of patients with at least one TEAE
- All treatment-emergent SAEs by primary SOC, showing number (%) of patients with at least one TEAE, sorted by internationally agreed order of primary SOC

# Analysis of all treatment-emergent adverse event(s) leading to treatment discontinuation

- All TEAEs leading to treatment discontinuation, by primary SOC, HLGT, HLT, and PT, showing number (%) of patients sorted by SOC internationally agreed order. The other level (HLGT, HLT, PT) will be presented in an alphabetic order.
- All TEAEs leading to treatment discontinuation, by primary SOC and PT, showing number (%) of patients with at least one TEAE
- All TEAEs leading to treatment discontinuation, by primary SOC, showing number (%) of patients with at least one TEAE, sorted by internationally agreed order of primary SOC

# Analysis of all treatment-emergent adverse event(s) leading to dose reduction

• For the management of pre-defined laboratory abnormalities, sarilumab dose can be reduced to 150 mg q2w. All treatment-emergent adverse events leading to dose reduction, by primary SOC, HLGT, HLT and PT, showing the number (%) of patients, sorted by the sorting order defined above

# Analysis AESI

- Summaries of AESI defined by the search criteria:
  - All treatment-emergent AESIs, by AESI category and PT, showing number (%) of patients, sorted by decreasing incidence of PT within each AESI category.
  - Within each treatment-emergent AESI category, at a minimum the data display will include:
    - Overview summary
    - Treatment duration summary
    - Incidence by patient and by event

- Serious TEAEs
- TEAEs leading to treatment discontinuation
- TEAEs leading to death
- Possibly related TEAEs

#### 2.4.5.2 Deaths

The incidence of death will be generated on the safety populations.

- Number (%) of patients who died by study period (on-treatment, treatment residual, and post-treatment).
- Death in non-randomized patients or randomized but not treated patients.
- TEAE leading to death (death as an outcome on the AE CRF page as reported by the Investigator) by primary SOC and PT, showing number (%) of patients sorted by internationally agreed order of SOC and and decreasing frequency of PT within a SOC in the Sarilumab 200mg q2w treatment group.

Listings will be provided for all deaths with flags indicating during treatment or post-treatment status.

# 2.4.5.3 Analyses of laboratory variables

The summary statistics (including number, mean, median, SD, minimum and maximum) of all laboratory variables (central laboratory values and changes from baseline) will be calculated for each visit or study assessment (baseline, each post baseline time point, endpoint) by treatment group. This section will be organized by biological function as specified in Section 2.1.4.3.

In addition, for all laboratory parameters, the mean value and mean change from baseline at each scheduled visit during the treatment period will be plotted by treatment group.

The incidence of PCSAs (list provided in Appendix B) at any time during TEAE period will be summarized by biological function and treatment group whatever the baseline level and/or according to the following baseline status categories:

- Normal/missing
- Abnormal according to PCSA criterion or criteria

For lipids, the National Cholesterol Education Program Adult Treatment Panel III (NCEP ATPIII) classification will be used for the baseline.

The incidence of abnormal laboratory values at any time during the TEAE period will be summarized in shift tables by biological function and treatment group whatever the baseline level and/or according to the following baseline status categories:

Normal/Missing

- Abnormal high according to the normal range
- Abnormal low according to the normal range

Time to onset of the initial LDL-C elevation ( $\geq$ 4.1 mmol/L,  $\geq$ 4.9 mmol/L), time to onset of the initial total cholesterol elevation ( $\geq$ 6.2 mmol/L), time to onset of the initial Grade 3 or Grade 4 neutropenia (neutrophil count <1.0 Giga/L), time to onset of the initial platelet count <100 Giga/L, time to onset of the initial lymphocyte count <1.0 Giga/L, time to onset of the initial ALT elevation (>3 x ULN, >5 x ULN), time to onset of the initial AST elevation (>3 x ULN, >5 x ULN), and time to onset of initial total bilirubin >2 x ULN will be analyzed using Kaplan-Meier estimates, using the midpoint of the time interval between the first assessment showing the elevation and the previous assessment, presented by treatment group.

Listings will be provided with flags indicating the out of range values as well as the PCSA values.

# Neutrophils

The incidence of neutropenia by maximal grade (lowest absolute neutrophil count reported during the TEAE period) will be summarized. The 4 grades are defined as below:

- Grade 1: ≥1.5 Giga/L-LLN.
- Grade 2:  $\geq$ 1.0 Giga/L-<1.5 Giga/L.
- Grade 3:  $\geq$ 0.5 Giga/L-  $\leq$ 1.0 Giga/L.
- Grade 4: <0.5 Giga/L.

#### **Thrombocytopenia**

The incidence of thrombocytopenia by maximal grade (lowest platelet count reported during the TEAE period) as defined below will be summarized.

- ≥75 Giga/L-100 Giga/L.
- $\geq$ 50 Giga/L-<75 Giga/L.
- ≥25 Giga/L-<50 Giga/L.
- <25 Giga/L.

#### Hepatic disorders

The liver function tests, namely AST, ALT, ALP, and total bilirubin are used to assess possible drug-induced liver toxicity. The proportion of patients with PCSA values at any post-baseline visit by baseline status will be displayed by treatment group for each parameter. The proportion of patients with PCSA values at any post baseline visit may be displayed by duration of exposure for each treatment group.

A graph of distribution of peak values of ALT versus peak values of total bilirubin will also be presented. Note that the ALT and total bilirubin values are presented on a logarithmic scale. The

graph will be divided into 4 quadrants with a vertical line corresponding to 3x ULN for ALT and a horizontal line corresponding to 2x ULN for total bilirubin.

# 2.4.5.4 Analyses of vital sign variables

The summary statistics (including number, mean, median, SD, minimum, and maximum) of all vital signs variables (vital signs values and changes from baseline) will be calculated for each visit or study assessment (baseline, each post baseline time point, endpoint) by treatment group.

The incidence of PCSAs at any time during the TEAE period will be summarized by treatment group whatever the baseline level and/or according to the following baseline status categories:

- Normal/Missing
- Abnormal according to PCSA criterion or criteria

Listings will be provided with flags indicating the PCSA values.

# 2.4.6 Analyses of pharmacokinetic variables

All the PK analyses will be performed using the PK populations including only the sarilumab treated patients.

Serum concentrations of functional sarilumab will be summarized using descriptive statistics (including number, arithmetic and geometric means, SD, standard error of the mean, coefficient of variation, minimum, median, and maximum) for each visit. The samples will be considered non-eligible for these analyses if the previous dosing time is <11 days or >17 days before the sampling time for every other week regimens. Concentrations below the lower limit of quantification (LLOQ) will be set to zero for samples at baseline (i.e., predose at Week 0). Other post-treatment concentrations below LLOQ will be replaced by LLOQ/2. In addition, serum concentrations of functional sarilumab will be summarized using descriptive statistics mentioned above by immunogenicity status for each visit.

Listings of serum concentration will be provided for each individual patient. The listings include subject identification (ID), gender, age, first dose date, visit number, categorized time point (0 for trough level and 1 for pre-dose), date/time of previous dose, PK sampling date/time, duration since first dose (days), duration since previous dose (dd:hh), serum concentration (ng/mL).

# 2.4.7 Analyses of quality of life variables

Descriptive statistics including number of subjects, mean, median, SD, minimum, maximum will be provided by treatment groups for the value and change from baseline at each visit (baseline, Week 12, Week 24 and Week 52) for the 2 summary measures of SF-36 (physical component summary score and mental component summary score) and the 8 domains, the quantitative variables of EQ-5D-3L (visual analog scale and single index utility), FACIT-Fatigue, HAQ-DI (standardized score, pain score and patient global assessment) and MD-VAS. Analyses will be performed based on data as observed; no missing data will be imputed.

# 2.4.8 Analysis of immunogenicity endpoints

The following summary will be provided separately for ADA positive patients, ADA negative patients, patients with persistent ADA response, and patients with transient ADA responses.

#### ADA prevalence and titer

The following summary will be provided based on the ADA populations:

- Number (%) of patients with an ADA positive sample at baseline:
  - Number (%) of neutralizing antibody.
  - Number (%) of non-neutralizing antibody.
  - The summary statistics (including number, median, Q1, Q3, minimum and maximum) of the titer for the baseline ADA positive patients.
- Number (%) of patients with an ADA negative sample at baseline.

#### ADA incidence and titer

The following summary will be provided based on the ADA populations during TEAE period:

- Number (%) of ADA-negative patients.
- Number (%) of ADA-positive patients:
  - Number (%) of patients with neutralizing antibody.
  - Number (%) of patients with non-neutralizing antibody.
  - The summary statistics (including number, median, Q1, Q3, minimum, and maximum) of the peak post-baseline titer for all ADA-positive patients.
- Number (%) of treatment-emergent ADA-positive patients:
  - The summary statistics (including number, median, Q1, Q3, minimum, and maximum) of the peak post-baseline titer for treatment-emergent ADA-positive patients.
  - Number (%) of transient treatment-emergent ADA-positive patients:
    - Number (%) of patients with neutralizing antibody.
    - Number (%) of patients with non-neutralizing antibody.
  - Number (%) of persistent treatment-emergent ADA positive patients:
    - Number (%) of patients with neutralizing antibody.
    - Number (%) of patients with non-neutralizing antibody.
  - Number (%) of persistent treatment-emergent ADA positive patients because last sample was positive.
- Number (%) of treatment-boosted ADA positive patients:

- Number (%) of patients with neutralizing antibody.
- Number (%) of patients with non-neutralizing antibody.
- The summary statistics (including number, median, Q1, Q3, minimum, and maximum) of the peak post-baseline titer for all treatment-boosted ADA-positive patients.

In addition, number (%) of patients with ADA positive or negative response at each visit will be summarized by treatment group.

#### ADA and PK

By visit descriptive summary of functional sarilumab concentrations in serum will be provided by ADA patient classifications (positive or negative) for the sarilumab treatment groups.

#### 2.4.9 **DNA/RNA**

The DNA test is optional and patients need to sign a separate informed consent for DNA testing. Exploratory analysis of DNA/RNA will be addressed in a separate document by a separate biomarker analysis group.

#### 2.5 DATA HANDLING CONVENTIONS

#### 2.5.1 General conventions

The following formulas will be used for computations of parameters.

# Demographic formulas:

BMI is calculated as follows:

BMI = Weight in kg/(height<sup>2</sup> in meters).

#### 2.5.2 Data handling conventions for secondary efficacy variables

#### **GTI**

# General Considerations

For vital signs and laboratory data used together with the GTI CRF to derive the scoring the scheduled measurements at the time of the visit should generally be used, but if any of these are missing they can be replaced by the last available measurement in the corresponding time window for that parameter.

#### GTI missing domains

The missing lab measurement for any GTI domain at a visit will be imputed by last observation carried forward (LOCF) method, and missing medication information for Glucose, Blood Pressure

and Hyperlipidemia domains will be imputed as 'no change' in order to calculate the composite and cumulative GTI scores.

# 2.5.3 Missing data

For categorical variables, patients with missing data are not included in calculations of percentages unless otherwise specified. When relevant, the number of patients with missing data is presented.

# Handling of computation of treatment duration if investigational medicinal product end of treatment date is missing

For the calculation of the treatment duration, the date of the last dose of SC IMP is equal to the date of last administration reported on the SC IMP administration CRF page. If this date is missing, the exposure duration should be left as missing.

# Handling of medication missing/partial dates

No imputation of medication start/end dates or times will be performed. If a medication date or time is missing or partially missing and it cannot be determined whether it was taken prior or concomitantly, it will be considered a prior and concomitant medication.

# Handling of AEs with missing or partial date/time of onset

Missing or partial missing AE onset dates and times will be imputed so that if the partial AE onset date/time information does not indicate that the AE started prior to treatment or after the TEAE period, the AE will be classified as treatment-emergent. No imputation of AE end dates/times will be performed. These data imputations are for categorization purpose only and will not be used in listings. No imputation is planned for date/time of AE resolution.

# Handling of AEs when date and time of first investigational medicinal product administration is missing

When the date and time of the first IMP administration is missing, all AEs that occurred on or after the day of randomization should be considered as TEAE. The exposure duration should be kept as missing.

# Handling of missing relationship of adverse events to investigational medicinal product

If the assessment of the relationship to IMP is missing, then the relationship to IMP has to be assumed and the AE considered as such in the frequency tables of possibly related AEs, but no imputation should be done at the data level.

# Handling of missing severity of AEs

If the severity is missing for one of the treatment-emergent occurrences of an AE, the maximal severity on the remaining occurrences will be considered. If the severity is missing for all the occurrences a "missing" category will be added in summary table.

# Handling of PCSA

If a patient has a missing baseline he will be grouped in the category "normal/missing at baseline."

For PCSAs with 2 conditions, one based on a change from baseline value or a normal range and the other on a threshold value, with the first condition being missing, the PCSA will be based only on the second condition.

For a PCSA defined on a threshold and/or a normal range, this PCSA will be derived using this threshold if the normal range is missing; eg, for eosinophils the PCSA is > 0.5 GIGA/L or >ULN if ULN  $\ge 0.5$  GIGA/L. When ULN is missing, the value 0.5 should be used.

Measurements flagged as invalid by the laboratory will not be summarized or taken into account in the computation of PCSA values.

# 2.5.4 Windows for time points

Visit windows based on days relative to the first IMP dose will be used to map the efficacy, lab, vital signs, PK and ADA measurements to each scheduled visit (see Appendix H). The following rule will be applied when mapping the measurements to the visit:

- For the same parameter (i.e., efficacy, lab, or vital signs), if a patient has more than one measurement at different dates within the same visit window, the scheduled measurement that is closest to the target date will be used (in case of tie select the latest). If there is no scheduled measurement within the visit window, the unscheduled measurement that is closest to the target date will be used (in case of tie select the latest).
- When a patient has more than one measurement on the same parameter on the same date, then the one with the later/largest sample ID will be used.
- If there is no measurement for a given parameter in an analysis window, data will be considered missing for the corresponding visit.

#### 2.5.5 Unscheduled visits

Unscheduled visit measurements of laboratory parameters and vital signs will be used for computation of baseline, the last on-treatment value, analysis according to PCSA analysis, and the shift summaries for safety. They will also be included in the by-visit summaries if they are reallocated to scheduled visits.

#### 2.5.6 Remote Assessment

Due to the nature of the COVID-19 pandemic, related travel restrictions, and on-site visits limitations, some efficacy assessments and laboratory parameters have been taken remotely or locally. All the measurements will be used in the analyses.

# 2.5.7 Pooling of centers for statistical analyses

Countries are pooled by region: Western countries, South American and Rest of the world.

- Region 1 (Western countries): Australia, Belgium, Canada, Croatia, Denmark, Estonia, France, Germany, Hungary, Italy, Netherlands, Portugal, Slovenia, Spain, Sweden, Switzerland, United Kingdom, United States.
- Region 2 (South American): Argentina.
- Region 3 (Rest of the world): Russia, Israel.

# 2.5.8 Statistical technical issues

Not applicable.

# 3 INTERIM ANALYSIS

No interim analysis is planned for this study.

# 4 DATABASE LOCK

The database lock will occur approximately 4 weeks after the last patient has completed the EOS Visit.

# 5 SOFTWARE DOCUMENTATION

All summaries and statistical analyses will be generated using SAS version 9.2 or higher.

# 6 REFERENCES

- 1. J.H. Stone, K. Tuckwell, S. Dimonaco, et al. Trial of Tocilizumab in Giant-Cell Arteritis. The New England Journal of Medicine. 2017;377(4):317–328.
- 2. Eli M. Miloslavsky, Ray P. Naden, Johannes W.J. Bijlsma, et al. Development of a Glucocorticoid Toxicity Index (GTI) using multicriteria decision analysis. Annals of the rheumatic diseases. 2017;76(3):543–546.
- 3. EurolQol Group. EuroQol-a new facility for the measurement of health-related quality of life. Health Policy. 1990;16(3):199-208.

# 7 LIST OF APPENDICES

Appendix A: Study flow chart

Appendix B: Potentially clinically significant abnormalities (PCSA) criteria

Appendix C: Summary of statistical analyses

Appendix D: SF-36 V2 Scoring

Appendix E: FACIT-Fatigue scoring guidelines (Version 4)

Appendix F: SAS code for EQ-5D-3L index utility scoring

Appendix G SAS code for SF-36 scoring

Appendix H Visit windows based on day ranges

Appendix I Baseline glucocorticoid toxicity

# Appendix A Study flow chart

| VISIT | V1 | V2 | V3 | V4 | V5 | V6 | V7 | V8 | V9 | V10 | V11 | V12<br>(EOT) | V13 | V14 (EOS) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| DAY | D -42 to<br>D -1 | D1 | D15<br>(±3) | D29<br>(±3) | D57<br>(±3) | D85 (±3) | D113 (±3) | D141<br>(±3) | D169 (±3) | D225 (±3) | D281 (±3) | D365 (±3) | D407<br>(±3) | D532 (±3) |
| WEEK | | Wk 0 | Wk 2 | Wk 4 | Wk 8 | Wk 12 | Wk 16 | Wk 20 | Wk 24 | Wk 32 | Wk 40 | Wk 52 | Wk 58 | Wk 76 |
| Eligibility | | | | | | | | | | | | | | |
| Written informed consent | Х | | | | | | | | | | | | | |
| Inclusion/exclusion criteria <sup>a</sup> | Χa | Х | | | | | | | | | | | | |
| Patient demography | Х | | | | | | | | | | | | | |
| Medical/surgical/smoking/alcohol history | Х | | | | | | | | | | | | | |
| Prior medication history | Х | | | | | | | | | | | | | |
| Family cardiovascular history | Х | | | | | | | | | | | | | |
| Full physical examination | Х | | | | | | | | | | | Х | | |
| Targeted physical examination <sup>b</sup> | | Х | | | | Х | | | Х | | Х | | | |
| Confirm eligibility | | Х | | | | | | | | | | | | |
| Randomization | | Х | | | | | | | | | | | | |
| Call IRT | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | | Х |
| Treatment | | | | | | | | | | | | | | |
| Initial treatment kit assignment (IRT) | | Х | | | | | | | | | | | | |
| IMP administration <sup>C</sup> | | Х | Х | Х | Χ | Х | Х | Х | χď | χď | Xď | Х | | |
| Concomitant medication review | Х | Χ | Χ | Х | Χ | Х | Х | Χ | Х | Х | Х | Х | Х | Х |
| Dispense patient diary (for study medications) | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | | | |
| Compliance/review patient diary | | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | | |

| VISIT | V1 | V2 | V3 | V4 | V5 | V6 | V7 | V8 | V9 | V10 | V11 | V12<br>(EOT) | V13 | V14 (EOS) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| DAY | D -42 to<br>D -1 | D1 | D15<br>(±3) | D29<br>(±3) | D57<br>(±3) | D85 (±3) | D113 (±3) | D141<br>(±3) | D169 (±3) | D225 (±3) | D281 (±3) | D365 (±3) | D407<br>(±3) | D532 (±3) |
| WEEK | | Wk 0 | Wk 2 | Wk 4 | Wk 8 | Wk 12 | Wk 16 | Wk 20 | Wk 24 | Wk 32 | Wk 40 | Wk 52 | Wk 58 | Wk 76 |
| Vital signs | | | | | | | | | | | | | | |
| Temperature, heart rate, blood pressure | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Weight | Х | Х | | | | Х | | | Х | | Х | Х | | |
| Height | Х | | | | | | | | | | | | | |
| Efficacy | | | | | | | | | | | | | | |
| GCA clinical assessments (including disease flare) | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| PROs <sup>e</sup> | | Х | | | | Х | | | Х | | | Х | | |
| Physician Global Assessment (MD-VAS) | | Х | | | | Х | | | Х | | | Х | | |
| GTI Assessment (excluding Bone Density assessment) | | Х | | | | Х | | | Х | | Х | Х | | |
| Bone density assessment <sup>f</sup> | | Х | | | | | | | | | | Х | | |
| Safety | | | | | | | | | | | | | | |
| AE/SAE recording | | | | | | | | | | | | | | |
| Tuberculosis assessment | Х | Х | Х | Х | Х | Х | Х | Χ | Х | Х | Х | Х | Χ | |
| QuantiFERON® | Х | | | | | | | | | | | | | |
| Chest X-ray <sup>g</sup> | Х | | | | | | | | | | | | | |
| Laboratory testing | | | | | | | | | | | | | | |
| Hematology <sup>h</sup> | Х | Х | | Х | | Х | | | Х | | Х | Х | | |
| Chemistry <sup>i</sup> | Х | Х | | Х | | Х | | | Х | | Х | Х | | |
| ANA | | Х | | | | | | | | | | Х | | |

| VISIT | V1 | V2 | V3 | V4 | V5 | V6 | V7 | V8 | V9 | V10 | V11 | V12<br>(EOT) | V13 | V14 (EOS) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| DAY | D -42 to<br>D -1 | D1 | D15<br>(±3) | D29<br>(±3) | D57<br>(±3) | D85 (±3) | D113 (±3) | D141<br>(±3) | D169 (±3) | D225 (±3) | D281 (±3) | D365 (±3) | D407<br>(±3) | D532 (±3) |
| WEEK | | Wk 0 | Wk 2 | Wk 4 | Wk 8 | Wk 12 | Wk 16 | Wk 20 | Wk 24 | Wk 32 | Wk 40 | Wk 52 | Wk 58 | Wk 76 |
| Fasting lipids <sup>j, k</sup> /fasting glucose, fasting insulin <sup>j</sup> | Х | | | Х | | Х | | | Х | | Х | Х | | |
| HbA1c | Х | | | Х | | Х | | | Х | | Х | Х | | |
| CRP <sup>I</sup> | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | | |
| ESR <sup>I</sup> | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | | |
| Urinalysis <sup>m</sup> | Х | | | | | | | | | | | | | |
| Virology <sup>n</sup> | Х | | | | | | | | | | | | | |
| Serum pregnancy test <sup>0</sup> | Х | | | | | | | | | | | | | |
| Urine pregnancy test <sup>0</sup> | | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х | | |
| 12-lead ECG | Х | | | | | | | | | | | | | |
| Serum sarilumab <sup>j</sup> | | Х | Х | Х | | Х | Х | | χ <mark>ρ</mark> | | | Х | Х | |
| Anti-drug antibody <sup>j</sup> | | Х | | | | Х | | | Х | | | Х | Х | |
| Genotyping and biomarkers <sup>j</sup> , | | | | | | | | | | | | | | |
| Biomarkers-IL-6 and sIL-6R | | Х | Х | | | Х | | | Х | | | Х | | |
| Blood for circulating immune cell ${\bf phenotyping}^{\it q}$ | | Х | | Х | | | | | Х | | | | | |
| Future Use of Samples for Circulating proteins (serum/ plasma) <sup>r</sup> (optional) | | Х | Х | | | Х | | | Х | | | Х | | |

| VISIT | V1 | V2 | V3 | V4 | V5 | V6 | V7 | V8 | V9 | V10 | V11 | V12<br>(EOT) | V13 | V14 (EOS) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| DAY | D -42 to<br>D -1 | D1 | D15<br>(±3) | D29<br>(±3) | D57<br>(±3) | D85 (±3) | D113 (±3) | D141<br>(±3) | D169 (±3) | D225 (±3) | D281 (±3) | D365 (±3) | D407<br>(±3) | D532 (±3) |
| WEEK | | Wk 0 | Wk 2 | Wk 4 | Wk 8 | Wk 12 | Wk 16 | Wk 20 | Wk 24 | Wk 32 | Wk 40 | Wk 52 | Wk 58 | Wk 76 |
| DNA <sup>S</sup> (optional) | | X | | | | | | | | | | | | |
| RNA <sup>S</sup> (optional) | | Х | Х | | | | | | | | | | | |

AE = Adverse event; ANA = Antinuclear antibodies; CRP = C-reactive protein; D = Day; DNA = Deoxyribonucleic acid; ECG = Electrocardiogram; EOT = End of treatment; EOS = End of study; EQ-5D-3L = EuroQol five-dimensional three-level questionnaire; ESR = Erythrocyte sedimentation rate; FACIT-Fatigue = Functional assessment of chronic illness therapy fatigue scale; GCA = Giant cell arteritis; GTI = Glucocorticoid toxicity index; HAQ-DI = Health assessment questionnaire disability index; HbA1c = Hemoglobin A1c; HBsAg = Hepatitis B surface antigen; HBcore Ab = Hepatitis B core antibodies; HCV = Hepatitis C virus; IL = Interleukin; IMP = Investigational medicinal product; IRT = Interactive response technology; MD-VAS = Physician global assessment of disease activity - visual analog scale; MRI = Magnetic resonance imaging; Pain VAS = Pain visual analog scale; PROs = Patient reported outcomes; Pt-VAS = Patient global assessment of disease activity - visual analog scale; RNA = Ribonucleic acid; SAE = Serious adverse event; SF-36v2 = Short form 36 version 2; TB = Tuberculosis; V = Visit; Wk = Week.

- a If ultrasound is being used as a diagnostic tool of GCA, the image needs to be submitted to the central reader for confirmation of eligibility.
- b Targeted physical examination: head, eyes, ears, neck and throat, skin, respiratory, cardiovascular, neurologic, lymphatic examinations and abdominal examination.
- c Last administration of sarilumab is at Week 50.
- d Where the visit interval exceeds 4 weeks, interim shipments of IMP to patients home may be performed using direct to patient (DTP) shipping (according to local regulations and logistics), in order to provide the patient with only 4 weeks IMP at a time in order to minimize compliance errors.
- e Patient Reported Outcomes include EQ-5D-3L, FACIT-Fatique, SF-36v2, HAQ-DI (including Pain VAS and Pt-VAS).
- f Bone mineral density assessment must be performed during baseline if not already available within 12 weeks prior to screening visit. A ±2 week time window is allowed at baseline visit and -2 week time window is allowed at EOT visit.
- g Posterior-Anterior chest X-ray must be performed during screening if not already available within 12 weeks prior to screening visit.

  A standard PA chest X-ray (lateral view is also recommended but not required) is required during the screening period if no chest imaging (X-ray, Computed Tomography [CT], MRI) is available within the previous 12 weeks of V1 that clearly documents the exclusion of TB (or >12 weeks, if appropriate according to local guidelines and requirements for screening of active TB). In countries for which a specific approval procedure for the X-ray is required by a different committee than the local ethics committee/Institutional review board (EC/IRB), a chest MRI between V1 and V2 can be performed.
- h Hematology (blood to be drawn before drug administration): Hemoglobin, hematocrit, red blood cell (RBC) count and morphology (if RBC count is abnormal), white blood cell (WBC) differential, platelet count, absolute neutrophil count (ANC).
- i Chemistry(blood to be drawn before drug administration): Sodium, potassium, chloride, bicarbonate, blood urea nitrogen (BUN), creatinine and creatinine clearance, calcium, phosphate, total protein, albumin, alanine aminotransferase (ALT) (SGPT), aspartate aminotransferase (AST) (SGOT), alkaline phosphatase (ALP), total bilirubin, conjugated bilirubin, unconjugated bilirubin, lactate dehydrogenase (LDH), uric acid.
- i Blood to be drawn before drug administration.
- k Lipids: Triglycerides (TG), total cholesterol, high density lipoprotein (HDL) cholesterol, low density lipoprotein (LDL) cholesterol.
- I CRP and ESR results will be blinded to Investigator (except screening and baseline). ESR kits will be provided by the central laboratory while the test will be performed locally at the site, results will be blinded to Investigator and staff directly involved in management of study patient, except safety assessor.
- m Urinalysis dipstick: specific gravity, pH, glucose, ketones, blood, protein, nitrite, leukocytes, urobilinogen and bilirubin. If any parameter on the dipstick is abnormal, a urine sample should be sent to the central laboratory for testing. If positive for proteins, microscopic analysis is performed by central laboratory.
- n Human immunodeficiency virus antibodies (a separate local Informed Consent may need to be obtained if applicable); Hepatitis B: HBsAg, total HB core Ab, Hep B Surface Antibody, and Hep B viral DNA (if necessary); Hepatitis C: HCV-antibodies.

Statistical Analysis Plan 08-Jan-2021 SAR153191-EFC15068 - sarilumab Version number: 1

- o In women of child-bearing potential.
- p Additional sample is to be drawn 4-7 days after Wk 24 dosing.
- q Immune cell phenotyping may be performed in only a subset of patients as determined by IRT system.
- r Future use Samples (for consented patients only).
- s Pharmacogenetic Research Informed Consent for collecting and sequencing DNA and RNA samples has to be obtained before any sampling. One DNA (at baseline) and RNA sample (predose) for sequencing sampling time point at baseline and V3 are needed.

# Appendix B Potentially clinically significant abnormalities (PCSA) criteria

# CRITERIA for POTENTIALLY CLINICALLY SIGNIFICANT ABNORMALITIES

for phase 2/3 studies (oncology excepted)

| Parameter | PCSA | Comments |
|---|---|---|
| Clinical Chemist | ry | |
| ALT | By distribution analysis: | Enzymes activities must be expressed in ULN, not in |
| | >3 ULN | IU/L. |
| | >5 ULN | Concept paper on DILI – FDA draft Guidance Oct 2007. |
| | >10 ULN | Internal DILI WG Oct 2008. |
| | >20 ULN | Categories are cumulative. |
| | Additional analysis*: | First row is mandatory. Rows following one |
| | >1 – 1.5 ULN | mentioning zero can be deleted. |
| | >1.5 – 3 ULN | |
| | >3 - 5 ULN | |
| | >5 – 8 ULN | |
| | > 8 ULN | |
| AST | By distribution analysis: | Enzymes activities must be expressed in ULN, not in |
| | >3 ULN | IU/L. |
| | >5 ULN | Concept paper on DILI – FDA draft Guidance Oct 2007. |
| | >10 ULN | Internal DILI WG Oct 2008. |
| | >20 ULN | Categories are cumulative |
| | Additional analysis*: | First row is mandatory. Rows following one |
| | >1 – 1.5 ULN | mentioning zero can be deleted. |
| | >1.5 – 3 ULN | |
| | >3 - 5 ULN | |
| | >5 – 8 ULN | |
| | > 8 ULN | |

for phase 2/3 studies (oncology excepted)

| Parameter | PCSA | Comments |
|---|---|---|
| Alkaline Phosphatase | >1.5 ULN | Enzymes activities must be expressed in ULN, not in IU/L. |
| | | Concept paper on DILI – FDA draft Guidance Oct 2007. |
| | | Internal DILI WG Oct 2008. |
| Total Bilirubin | >1.5 ULN | Must be expressed in ULN, not in µmol/L or mg/L. |
| | >2 ULN | Concept paper on DILI – FDA draft Guidance Oct 2007. |
| | | Internal DILI WG Oct 2008. |
| | | Categories are cumulative. |
| | | First row is mandatory. Rows following one mentioning zero can be deleted. |
| Conjugated Bilirubin | >35% Total Bilirubin and TBILI>1.5 ULN | Conjugated bilirubin dosed on a case-by-case basis. |
| | Additional analysis*: | PCSA to be retrieved manually |
| | >1.5 ULN | |
| | >2 ULN | |
| Unconjugated bilirubin | Additional analysis*: | Must be expressed in ULN, not in µmol/L or mg/L. |
| | >1.5 ULN | Categories are cumulative. |
| | >2 ULN | |
| ALT and Total Bilirubin | ALT>3 ULN and TBILI>2 ULN | Concept paper on DILI – FDA draft Guidance Oct 2007. |
| | | Internal DILI WG Oct 2008. |
| | | To be counted within a same treatment phase, whatever the interval between measurement. |

for phase 2/3 studies (oncology excepted)

| Parameter | PCSA | Comments |
|---|---|---|
| CPK** | >3 ULN | FDA Feb 2005. |
| | >10 ULN | Am J Cardiol April 2006. |
| | | Categories are cumulative. |
| | | First row is mandatory. Rows following one mentioning zero can be deleted. |
| Creatinine | ≥150 µmol/L (Adults) | Benichou C., 1994. |
| | ≥30% change from baseline | |
| | ≥100% change from baseline | |
| CLcr (mL/min) | <15 (end stage renal disease) | FDA draft Guidance 2010 |
| (Estimated creatinine | ≥15 - <30 (severe decrease in GFR) | Pharmacokinetics in patients with impaired renal |
| clearance based on the Cokcroft-Gault equation) | ≥30 - < 60 (moderate decrease in GFR) | function-study design, data analysis, and impa<br>dosing and labeling |
| ookoron-Gaan equation) | ≥60 - <90 (mild decrease in GFR) | dosing and laboring |
| | ≥ 90 (normal GFR) | |
| eGFR** (mL/min/1.73m2) | <15 (end stage renal disease) | FDA draft Guidance 2010 |
| (Estimate of GFR based | ≥15 - <30 (severe decrease in GFR) | Pharmacokinetics in patients with impaired renal |
| on an MDRD equation) | ≥30 - < 60 (moderate decrease in GFR) | function-study design, data analysis, and impact on dosing and labeling |
| | ≥60 - <90 (mild decrease in GFR) | dosing and laboring |
| | ≥ 90 (normal GFR) | |
| Uric Acid | | Harrison- Principles of internal Medicine 17th Ed., |
| Hyperuricemia | >408 µmol/L | 2008. |
| Hypouricemia | <120 µmol/L | |
| Blood Urea Nitrogen | ≥17 mmol/L | |
| Chloride | <80 mmol/L | |
| | >115 mmol/L | |
| Sodium | ≤129 mmol/L | |
| | ≥160 mmol/L | |

for phase 2/3 studies (oncology excepted)

| Parameter | PCSA | Comments |
|---|---|---|
| Potassium | <3 mmol/L | FDA Feb 2005. |
| | ≥5.5 mmol/L | |
| Total Cholesterol | ≥7.74 mmol/L | Threshold for therapeutic intervention. |
| | ≥6.2 mmol/L* | |
| LDL | ≥4.1 mmol/L* | |
| | ≥4.9 mmol/L | |
| Triglycerides | ≥4.6 mmol/L | Threshold for therapeutic intervention. |
| | ≥5.6 mmol/L* | |
| Lipasemia** | ≥3 ULN | |
| Amylasemia** | ≥3 ULN | |
| Glucose | | |
| Hypoglycaemia | ≤3.9 mmol/L and <lln< td=""><td>ADA May 2005.</td></lln<> | ADA May 2005. |
| Hyperglycaemia | ≥11.1 mmol/L (unfasted); ≥7 mmol/L (fasted) | ADA Jan 2008. |
| HbA1c | >8% | |
| Albumin | ≤25 g/L | |
| CRP | >2 ULN or >10 mg/L (if ULN not provided) | FDA Sept 2005. |
| Hematology | | |
| WBC | <3.0 Giga/L (Non-Black); <2.0 Giga/L (Black) | Increase in WBC: not relevant. |
| | ≥16.0 Giga/L | To be interpreted only if no differential count available. |
| Lymphocytes | <0.5 Giga/L* | |
| | ≥0.5 Giga/L - LLN* | |
| | >4.0 Giga/L | |
| Neutrophils | <1.5 Giga/L (Non-Black);<1.0 Giga/L (Black) | International Consensus meeting on drug-induced |
| | <1.0 Giga/L* | blood cytopenias, 1991. |
| | | FDA criteria. |

for phase 2/3 studies (oncology excepted)

| Parameter | PCSA | Comments |
|---|---|---|
| Monocytes | >0.7 Giga/L | |
| Basophils | >0.1 Giga/L | |
| Eosinophils | >0.5 Giga/L or >ULN (if ULN≥0.5 Giga/L) | Harrison- Principles of internal Medicine 17 <sup>th</sup> Ed., 2008. |
| Hemoglobin | ≤115 g/L (Male); ≤95 g/L (Female) | Criteria based upon decrease from baseline are |
| | ≥185 g/L (Male); ≥165 g/L (Female) | more relevant than based on absolute value. Ot categories for decrease from baseline can be us (≥30 g/L, ≥40 g/L, ≥50 g/L). |
| | Decrease from Baseline ≥20 g/L | |
| Hematocrit | ≤0.37 v/v (Male) ; ≤0.32 v/v (Female) | |
| | ≥0.55 v/v (Male) ; ≥0.5 v/v (Female) | |
| RBC | ≥6 Tera/L | Unless specifically required for particular drug development, the analysis is redundant with that of Hb. |
| | | Otherwise, consider FDA criteria. |
| Platelets | < 50 Giga/L* | International Consensus meeting on drug-induced |
| | ≥ 50 - 100 Giga/L* | blood cytopenias, 1991. |
| | ≥700 Giga/L | |
| Urinalysis | | |
| рН | ≤4.6 | |
| | ≥8 | |
| Vital signs | | |
| HR | ≤50 bpm and decrease from baseline ≥20 bpm | To be applied for all positions (including missing) |
| | ≥120 bpm and increase from baseline≥20 bpm | except STANDING. |
| SBP | ≤95 mmHg and decrease from baseline ≥20mmHg | To be applied for all positions (including missing) |
| | ≥160 mmHg and increase from baseline ≥20 mmHg | except STANDING. |
| DBP | ≤45 mmHg and decrease from baseline ≥10 mmHg | To be applied for all positions (including missing) |
| | ≥110 mmHg and increase from baseline ≥10 mmHg | except STANDING. |

for phase 2/3 studies (oncology excepted)

| Parameter | PCSA | Comments |
|-----------------------|----------------------------|---------------|
| Orthostatic Hypotensi | on | |
| Orthostatic SDB | | |
| Orthostatic DBP | ≤-20 mmHg | |
| | ≤-10 mmHg | |
| Weight | ≥5% increase from baseline | FDA Feb 2007. |
| | ≥5% decrease from baseline | |

08-Jan-2021 Version number: 1

# Appendix C Summary of statistical analyses

| | Analysis | | Statistical | Supportive | Subgroup | Other |
|---|---|---|---|---|---|---|
| Endpoint | Population | Primary Analysis | Method | Analysis* | Analysis* | Analyses* |
| Primary Endpoint | | | | | | |
| Patients who achieved sustained remission at Week 52 | ITT | Proportion of patients achieving sustained remission at Week 52 | CMH test stratified<br>by baseline<br>prednisone dose for<br>combined groups,<br>and descriptive<br>analysis for non-<br>combined groups. | 1) Sensitivity analysis;2) Analysis excluding patients who prematurely withdraw from the study due to early termination of the study | No | No |
| Additional endpoint:<br>Patients who achieved<br>sustained remission at<br>Week 24 | ITT | Proportion of patients achieving sustained remission at Week 24 | CMH test stratified<br>by baseline<br>prednisone dose for<br>combined groups,<br>and descriptive<br>analysis for non-<br>combined groups | Sensitivity analysis | No | No |
| Secondary Endpoints | | | | | | |
| Patients who achieved of disease remission by Week 12 | ITT | Proportion of patients who achieved of disease remission by Week 12 | Descriptive | No | No | No |
| Patients who have absence<br>of disease flare from Week<br>12 through Week 24 and<br>Week 52 | ITT | Proportion of patients who have absence of disease flare from Week 12 through Week 24 and Week 52 | Descriptive | No | No | No |
| Patients who have normalization of CRP (decrease to <10 mg/L) with sustained normalization from Week | ITT | Proportion of patients who have<br>normalization of CRP (decrease to<br><10 mg/L) with sustained<br>normalization from Week 12 through<br>Week 24 and Week 52 | Descriptive | No | No | No |

| | Analysis | | Statistical | Supportive | Subgroup | Other |
|---|---|---|---|---|---|---|
| Endpoint | Population | Primary Analysis | Method | Analysis* | Analysis* | Analyses* |
| 12 through Week 24 and Week 52 | | | | | | |
| Patients who successfully<br>adhere to the prednisone<br>taper from Week 12<br>through Week 24 and Week<br>52 | ITT | Proportion of patients who successfully adhere to the prednisone taper from Week 12 through Week 24 and Week 52 | Descriptive | No | No | No |
| Total cumulative prednisone (or equivalent) dose | ITT | Total cumulative prednisone (or equivalent) dose over 52-week treatment period | Descriptive | No | No | No |
| Time to the first GCA flare<br>after clinical remission up to<br>Week 52 | ITT | Time (from randomization) to the first<br>GCA flare after clinical remission up to<br>Week 52 | Kaplan-Meier estimates and Cox proportional hazards model for combined groups, and descriptive analysis for non-combined groups. | No | No | No |
| Total composite GTI total score | ITT | Cumulative GTI scores (CWS and AIS) at Week 24 and Week 52 | Descriptive by 4 treatment groups; and analysis of covariance (ANCOVA) model for combined groups. | No | No | Summaries of domain<br>specific scores and<br>specific list events at<br>Week 12, 24, 40 and 52. |
| Safety | | | | | | |
| Adverse Events | Safety | Follow safety guidelines | Descriptive | No | No | No |
| Laboratory | Safety | Follow safety guidelines | Descriptive | No | No | No |
| Vital signs and ECGs | Safety | Follow safety guidelines | Descriptive | No | No | No |

Statistical Analysis Plan SAR153191-EFC15068 - sarilumab 08-Jan-2021 Version number: 1

| Analysis | | | Statistical | Supportive | Subgroup | Other |
|---|---|---|---|---|---|---|
| Endpoint | Population | Primary Analysis | Method | Analysis* | Analysis* | Analyses* |
| PK | | | | | | |
| Sarilumab serum concentration | PK | By visit | Descriptive | No | No | No |
| Immunogenicity | | | | | | |
| ADA positive patients | ADA | NA | Descriptive | No | No | No |
| ADA negative patients | ADA | NA | Descriptive | No | No | No |
| Persistent ADA response | ADA | NA | Descriptive | No | No | No |
| Transient ADA response | ADA | NA | Descriptive | No | No | No |

# Appendix D SF-36 V2 Scoring

#### **General Scoring information**

Items and scales are scored in 3 steps:

- Step 1. Item recoding, for the 10 items that require recoding,
- Step 2. Computing scale scores by summing across items in the same scale (raw scale scores); and,
- Step 3. Transforming raw scale scores to a 0-100 scale (transformed scale).

# Item recoding

- All 36 items should be checked for out-of-range values prior to assigning the final item value. All out-of-range values should be recoded as missing data.
- The following tables show the recoding of response choice.

# How to treat missing data

A scale score is calculated if a respondent answered at least half of the items in a multi-item scale (or half plus one in the case of scales with an odd number of items).

The recommended algorithm substitutes a person-specific estimate for any missing item when the respondent answered at least 50 percent of the items in a scale. A psychometrically sound estimate is the average score, across completed items in the same scale, for that respondent. For example, if a respondent leaves one item in the 5-item mental Health scale blank, substitute the respondent's average score (across the 4 completed mental health items) for that one item. When estimating the respondent's average score, use the respondent's final item values.

#### **Computing raw scale scores**

After item recoding, including handling of missing data, a raw score is computed for each scale. This score is a simple algebraic sum of responses for all items in that scale.

If the respondent answered at least 50% of the items in a multi-items scale, the score can be calculated. If the respondent did not answer at least 50% of the items, the score for that scale should be set to missing.

# Transformation of the scale scores

The next step involves transforming each raw score to a 0 to 100 scale using the following formula:

Transformed scale = [(actual raw score – lowest possible raw score) / possible raw score range] x 100

This transformation converts the lowest and highest possible scores to zero and 100, respectively.

Table 8 - SF-36 V2 raw scores of eight domains

| Scale | Lowest and highest possible raw scores | Possible raw score range |
|---|---|---|
| Physical Functioning | 10,30 | 20 |
| Role-Physical | 4,20 | 16 |
| Bodily pain | 2,12 | 10 |
| General health | 5,25 | 20 |
| Vitality | 4,20 | 16 |
| Social Functioning | 2,10 | 8 |
| Role-Emotional | 3,15 | 12 |
| Mental Health | 5,25 | 20 |
## Appendix E FACIT-fatigue scoring guidelines (version 4)

Instructions:\* 1. Record answers in "item response" column. If missing, mark with an X

- 2. Perform reversals as indicated, and sum individual items to obtain a score.
- 3. Multiply the sum of the item scores by the number of items in the subscale, then divide by the number of items answered. This produces the subscale score.
- 4. The higher the score, the better the QOL.

| Subscale | <u>Item Code</u> | Reverse item? | <u>Item response</u> | Item Score |
|---|---|---|---|---|
| FATIGUE | HI7 | 4 - | | = |
| SUBSCALE | HI12 | 4 - | | = |
| | An1 | 4 - | | = |
| | An2 | 4 - | | = |
| | An3 | 4 - | | = |
| | An4 | 4 - | | = |
| | An5 | 0 + | | = |
| | An7 | 0 + | | = |
| | An8 | 4 - | | = |
| | An12 | 4 - | | = |
| | An14 | 4 - | | = |
| | An15 | 4 - | | = |
| | An16 | 4 - | | = |

Sum individual item scores:\_\_\_\_

Multiply by 13: \_\_\_\_\_

Divide by number of items answered: \_\_\_\_\_=Fatigue Subscale score

<sup>\*</sup>For guidelines on handling missing data and scoring options, please refer to the Administration and Scoring Guidelines in the manual or on-line at www.facit.org.

## Appendix F SAS code for EQ-5D-3L index utility scoring

```
/*----*/;
/* Aim : Derive the EQ5-D index (utility) */;
/* Source for the algorithm : scoring EQ-5D health states (Rosalind Rabin */;
/* (cf. G:\ HE\PRO questionnaire\EQ5D\scoring\YorkTariffx.doc) */;
/* Note: UK based population (Dolan, 1997) */;
/* Author : Elisheva Smadja */;
/*----*/;
data EUROQOL; set temp;
profil= (10000*eqq1cd)+(1000*eqq2cd)+(100*eqq3cd)+(10*eqq4cd)+eqq5cd;
eq5d=1;
*********Mobility*********;
if eqq1cd=2 then eq5d=eq5d-0.069;
if eqq1cd=3 then eq5d=eq5d-0.314;
*******Self-care*******;
if egg2cd=2 then eg5d=eg5d-0.104;
if egg2cd=3 then eg5d=eg5d-0.214;
******Usual activities****;
if eqq3cd=2 then eq5d=eq5d-0.036;
if eqq3cd=3 then eq5d=eq5d-0.094;
****Pain/discomfort****;
if eqq4cd=2 then eq5d=eq5d-0.123;
if eqq4cd=3 then eq5d=eq5d-0.386;
*****Anxiety/depression****;
if eqq5cd=2 then eq5d=eq5d-0.071;
if eqq5cd=3 then eq5d=eq5d-0.236;
if (eqq1cd ne 1 or eqq2cd ne 1 or eqq3cd ne 1 or eqq4cd ne 1 or eqq5cd ne 1)
then eq5d=eq5d-0.081;
if (eqq1cd=3 or eqq2cd=3 or eqq3cd=3 or eqq4cd=3 or eqq5cd=3)
then eq5d=eq5d-0.269;
if (eqq1cd=. or eqq2cd=. or eqq3cd=. or eqq4cd=. or eqq5cd=.)
then eq5d=.;
run;
```

## Appendix G SAS code for SF-36 scoring

```
******************
 PROGRAM: SF36 V2
* PURPOSE: SAS SCORING PROGRAM FOR THE SF-36 VERSION2
***********************
*************************
            STEP 1: INPUT DATA
*************************
DATA SF36DATA;
INFILE IN;
INPUT ID $ 1-3
    @ 5 (GH1 HT PF01-PF10 RP1-RP4 RE1-RE3 SF1
    BP1-BP2 VT1 MH1 MH2 MH3 VT2 MH4 VT3 MH5
    VT4 SF2 GH2 GH3 GH4 GH5) (1.);
RUN;
***********************
           STEP 2: SF-36 SCALE CONSTRUCTION
************************
USING THE SAS DATASET CREATED IN PART 1, CHANGE OUT-OF-RANGE
 VALUES TO MISSING FOR EACH ITEM. RECODE AND RECALIBRATE ITEMS
* AS NEEDED. AN 'R' PREFIX MEANS THE VARIABLE IS RECODED.
*********************
DATA SF36SCAL;
 SET SF36DATA;
***************
 THE SF-36 PHYSICAL FUNCTIONING INDEX.
 ALL ITEMS ARE POSITIVELY SCORED -- THE HIGHER THE ITEM
 VALUE, THE BETTER THE PHYSICAL HEALTH.
 THIS SCALE IS POSITIVELY SCORED.
* THE HIGHER THE SCORE THE BETTER THE PHYSICAL FUNCTIONING.
**********************
ARRAY PFI(10) PF01-PF10;
DO I = 1 TO 10;
 IF PFI(I) < 1 OR PFI(I) > 3 THEN PFI(I) = .;
END;
PFNUM = N(OF PF01-PF10);
PFMEAN = MEAN(OF PF01-PF10);
DO I = 1 TO 10;
IF PFI(I) = . THEN PFI(I) = PFMEAN;
```

```
END;
IF PFNUM GE 5 THEN RAWPF = SUM(OF PF01-PF10);
PF = ((RAWPF - 10)/(30-10)) * 100;
LABEL PF = 'SF-36 PHYSICAL FUNCTIONING (0-100)'
      RAWPF = 'RAW SF-36 PHYSICAL FUNCTIONING';
*****************
* THE SF-36 ROLE-PHYSICAL INDEX.
  ALL ITEMS ARE POSITIVELY SCORED -- THE HIGHER THE ITEM VALUE,
  THE BETTER THE ROLE-PHYSICAL FUNCTIONING.
  THIS SCALE IS POSITIVELY SCORED.
* THE HIGHER THE SCORE THE BETTER THE ROLE-PHYSICAL.
********************
ARRAY RPA(4) RP1-RP4;
DO I = 1 TO 4;
  IF RPA(I) < 1 OR RPA(I) > 5 THEN RPA(I) = .;
END;
ROLPNUM = N(OF RP1-RP4);
ROLPMEAN = MEAN(OF RP1-RP4);
DO I = 1 TO 4;
  IF RPA(I) = . THEN RPA(I) = ROLPMEAN;
END;
IF ROLPNUM GE 2 THEN RAWRP = SUM(OF RP1-RP4);
RP = ((RAWRP - 4)/(20-4)) * 100;
LABEL RP = 'SF-36 ROLE-PHYSICAL (0-100)'
     RAWRP = 'RAW SF-36 ROLE-PHYSICAL';
******************
  THE SF-36 PAIN ITEMS.
  ITEM RECODING DEPENDS ON WHETHER BOTH PAIN1 AND PAIN2
  ARE ANSWERED OR WHETHER ONE OF THE ITEMS HAS MISSING DATA.
  AFTER RECODING, ALL ITEMS ARE POSITIVELY SCORED -- THE HIGHER
  THE SCORE, THE LESS PAIN (OR THE MORE FREEDOM FROM PAIN).
   THIS SCALE IS POSITIVELY SCORED. THE HIGHER THE
   SCORE THE LESS PAIN OR THE MORE FREEDOM FROM PAIN.
*********************
IF BP1 < 1 OR BP1 > 6 THEN BP1 = .;
IF BP2 < 1 OR BP2 > 5 THEN BP2 = .;
* RECODES IF NEITHER BP1 OR BP2 HAS A MISSING VALUE;
IF BP1 NE . AND BP2 NE . THEN DO;
  IF BP1 = 1 THEN RBP1 = 6;
```

```
IF BP1 = 2 THEN RBP1 = 5.4;
   IF BP1 = 3 THEN RBP1 = 4.2;
   IF BP1 = 4 THEN RBP1 = 3.1;
   IF BP1 = 5 THEN RBP1 = 2.2;
  IF BP1 = 6 THEN RBP1 = 1;
  IF BP2 = 1 AND BP1 = 1 THEN RBP2 = 6;
   IF BP2 = 1 AND 2 LE BP1 LE 6 THEN RBP2 = 5;
  IF BP2 = 2 AND 1 LE BP1 LE 6 THEN RBP2 = 4;
  IF BP2 = 3 AND 1 LE BP1 LE 6 THEN RBP2 = 3;
  IF BP2 = 4 AND 1 LE BP1 LE 6 THEN RBP2 = 2;
  IF BP2 = 5 AND 1 LE BP1 LE 6 THEN RBP2 = 1;
END;
* RECODES IF BP1 IS NOT MISSING AND BP2 IS MISSING;
IF BP1 NE . AND BP2 = . THEN DO;
  IF BP1 = 1 THEN RBP1 = 6;
  IF BP1 = 2 THEN RBP1 = 5.4;
  IF BP1 = 3 THEN RBP1 = 4.2;
  IF BP1 = 4 THEN RBP1 = 3.1;
  IF BP1 = 5 THEN RBP1 = 2.2;
  IF BP1 = 6 THEN RBP1 = 1;
  RBP2 = RBP1;
END;
* RECODES IF BP1 IS MISSING AND BP2 IS NOT MISSING;
IF BP1 = . AND BP2 NE . THEN DO;
  IF BP2 = 1 THEN RBP2 = 6;
  IF BP2 = 2 THEN RBP2 = 4.75;
  IF BP2 = 3 THEN RBP2 = 3.5;
  IF BP2 = 4 THEN RBP2 = 2.25;
  IF BP2 = 5 THEN RBP2 = 1;
  RBP1 = RBP2;
END;
BPNUM = N(BP1, BP2);
IF BPNUM GE 1 THEN RAWBP = SUM(RBP1, RBP2);
BP = ((RAWBP - 2)/(12-2)) * 100;
LABEL BP = 'SF-36 PAIN INDEX (0-100)'
      RAWBP = 'RAW SF-36 PAIN INDEX';
************
  THE SF-36 GENERAL HEALTH PERCEPTIONS INDEX.
  REVERSE TWO ITEMS AND RECALIBRATE ONE ITEM. AFTER RECODING
  AND RECALIBRATION, ALL ITEMS ARE POSITIVELY SCORED -- THE
  HIGHER THE SCORE, THE BETTER THE PERCEIVED GENERAL HEALTH.
```

```
* THIS SCALE IS POSITIVELY SCORED.
* THE HIGHER THE SCORE THE BETTER THE HEALTH PERCEPTIONS.
************************
ARRAY GHP(5) GH1-GH5;
DO I = 1 TO 5;
 IF GHP(I) < 1 OR GHP(I) > 5 THEN GHP(I) = .;
END;
IF GH1 = 1 THEN RGH1 = 5;
IF GH1 = 2 THEN RGH1 = 4.4;
IF GH1 = 3 THEN RGH1 = 3.4;
IF GH1 = 4 THEN RGH1 = 2;
IF GH1 = 5 THEN RGH1 = 1;
RGH3 = 6 - GH3;
RGH5 = 6 - GH5;
GHNUM = N(GH1, GH2, GH3, GH4, GH5);
GHMEAN = MEAN(RGH1,GH2,RGH3,GH4,RGH5);
ARRAY RGH(5) RGH1 GH2 RGH3 GH4 RGH5;
DO I = 1 TO 5;
 IF RGH(I) = . THEN RGH(I) = GHMEAN;
END;
IF GHNUM GE 3 THEN RAWGH = SUM(RGH1, GH2, RGH3, GH4, RGH5);
GH = ((RAWGH - 5)/(25-5)) * 100;
LABEL GH = 'SF-36 GENERAL HEALTH PERCEPTIONS (0-100)'
      RAWGH = 'RAW SF-36 GENERAL HEALTH PERCEPTIONS';
******************
  THE SF-36 VITALITY ITEMS.
* REVERSE TWO ITEMS. AFTER ITEM REVERSAL, ALL ITEMS ARE
  POSITIVELY SCORED -- THE HIGHER THE SCORE, THE LESS THE FATIGUE
  AND THE GREATER THE ENERGY.
* THIS SCALE IS POSITIVELY SCORED.
* THE HIGHER THE SCORE THE GREATER THE VITALITY.
*************************************
ARRAY VI(4) VT1-VT4;
DO I = 1 TO 4;
 IF VI(I) < 1 OR VI(I) > 5 THEN VI(I) = .;
END;
RVT1 = 6-VT1;
RVT2 = 6-VT2;
VITNUM = N(VT1, VT2, VT3, VT4);
VITMEAN = MEAN(RVT1, RVT2, VT3, VT4);
```

```
ARRAY RVI(4) RVT1 RVT2 VT3 VT4;
DO I = 1 TO 4;
 IF RVI(I) = . THEN RVI(I) = VITMEAN;
END:
IF VITNUM GE 2 THEN RAWVT= SUM(RVT1,RVT2,VT3,VT4);
VT = ((RAWVT-4)/(20-4)) * 100;
LABEL VT = 'SF-36 VITALITY (0-100)'
     RAWVT = 'RAW SF-36 VITALITY';
***************
  THE SF-36 SOCIAL FUNCTIONING INDEX.
* REVERSE ONE ITEM SO THAT BOTH ITEMS ARE POSITIVELY SCORED --
  THE HIGHER THE SCORE, THE BETTER THE SOCIAL FUNCTIONING.
* THIS SCALE IS POSITIVELY SCORED.
* THE HIGHER THE SCORE THE BETTER THE SOCIAL FUNCTIONING.
******************
ARRAY SOC(2) SF1-SF2;
DO I = 1 TO 2;
  IF SOC(I) < 1 OR SOC(I) > 5 THEN SOC(I) = .;
END;
RSF1 = 6 - SF1;
SFNUM = N(SF1, SF2);
SFMEAN = MEAN(RSF1, SF2);
ARRAY RSF(2) RSF1 SF2;
DO I = 1 TO 2;
 IF RSF(I) = . THEN RSF(I) = SFMEAN;
END;
IF SFNUM GE 1 THEN RAWSF = SUM(RSF1, SF2);
SF = ((RAWSF - 2)/(10-2)) * 100;
LABEL SF = 'SF-36 SOCIAL FUNCTIONING (0-100)'
      RAWSF = 'RAW SF-36 SOCIAL FUNCTIONING';
******************
  THE SF-36 ROLE-EMOTIONAL INDEX.
  ALL ITEMS ARE POSITIVELY SCORED -- THE HIGHER THE ITEM VALUE,
  THE BETTER THE ROLE-EMOTIONAL FUNCTIONING.
  THIS SCALE IS POSITIVELY SCORED.
  THE HIGHER THE SCORE, THE BETTER THE ROLE-EMOTIONAL.
ARRAY RM(3) RE1-RE3;
```

```
DO I = 1 TO 3;
  IF RM(I) < 1 OR RM(I) > 5 THEN RM(I) = .;
END:
ROLMNUM = N(OF RE1-RE3);
ROLMMEAN = MEAN (OF RE1-RE3);
DO I = 1 TO 3;
  IF RM(I) = . THEN RM(I) = ROLMMEAN;
END:
IF ROLMNUM GE 2 THEN RAWRE = SUM(OF RE1-RE3);
RE = ((RAWRE - 3)/(15-3)) * 100;
LABEL RE = 'SF-36 ROLE-EMOTIONAL (0-100)'
      RAWRE = 'RAW SF-36 ROLE-EMOTIONAL';
**************
  THE SF-36 MENTAL HEALTH INDEX.
* REVERSE TWO ITEMS. AFTER ITEM REVERSAL, ALL ITEMS ARE
  POSITIVELY SCORED -- THE HIGHER THE SCORE, THE BETTER THE
  MENTAL HEALTH.
  THIS SCALE IS POSITIVELY SCORED.
* THE HIGHER THE SCORE THE BETTER THE MENTAL HEALTH.
*********************
ARRAY MHI(5) MH1-MH5;
DO I = 1 TO 5;
  IF MHI(I) < 1 OR MHI(I) > 5 THEN MHI(I)=.;
END:
RMH3 = 6-MH3;
RMH5 = 6-MH5;
MHNUM=N (MH1, MH2, MH3, MH4, MH5);
MHMEAN=MEAN (MH1, MH2, RMH3, MH4, RMH5);
ARRAY RMH(5) MH1 MH2 RMH3 MH4 RMH5;
DO I = 1 TO 5;
  IF RMH(I) = . THEN RMH(I) = MHMEAN;
END;
IF MHNUM GE 3 THEN RAWMH = SUM(MH1, MH2, RMH3, MH4, RMH5);
MH = ((RAWMH-5)/(25-5)) * 100;
LABEL MH = 'SF-36 MENTAL HEALTH INDEX (0-100)'
      RAWMH = 'RAW SF-36 MENTAL HEALTH INDEX';
*****************
* THE SF-36 HEALTH TRANSITION ITEM.
```

```
* THIS ITEM SHOULD BE ANALYZED AS CATEGORICAL DATA,
* PENDING FURTHER RESEARCH.
******************
IF HT < 1 OR HT > 5 THEN HT = .;
LABEL HT='RAW SF-36 HEALTH TRANSITION ITEM';
RUN:
**********************
           STEP 3: SF-36 SCALE CONSTRUCTION
DATA SF36INDX;
SET SF36SCAL;
********************
* purpose: create physical and mental health index scores
   standardized but not normalized
       and standard deviations calculated with vardef=wdf
*******************
/* NORM-BASED SCORING OF SF-36, STANDARD RECALL (4 WEEKS)
/* USING WEIGHTED MEANS AND SD'S FROM 1998 GENERAL US POPULATION
/* FROM COMBINED SAMPLES
*************
*****************
*CREATING SF-36 STANDARDIZED SCORES (0-100 Means/SD's from 1998 General
Population) *;
pf_z = (pf-83.29094)/23.75883;
rp z=(rp-82.50964)/25.52028;
bp z=(bp-71.32527)/23.66224;
gh z=(gh-70.84570)/20.97821;
 z=(vt-58.31411)/20.01923;
 z=(sf-84.30250)/22.91921;
re z=(re-87.39733)/21.43778;
mh z=(mh-74.98685)/17.75604;
*;
   COMPUTE SAMPLE RAW FACTOR SCORES
   Z SCORES ARE FROM ABOVE
                                       *;
   SCORING COEFFICIENTS ARE FROM U.S. GENERAL POPULATION *;
   FACTOR ANALYTIC SAMPLE N=2393: HAVE ALL EIGHT SCALES
****************
```

# Appendix H Visit windows based on day ranges

Visit windows based on days relative to the first IMP dose will be used to map (see Table 9).

Table 9 - Day range for each scheduled visit in the DB period for efficacy, lab, vital sign, PK and ADA summaries

| Visit Label | Target<br>Day | Schedule A <sup>a</sup> | Schedule B <sup>b</sup> | Schedule C <sup>C</sup> | Schedule D <sup>d</sup> | Schedule E <sup>e</sup> | Schedule F <sup>f</sup> | Schedule<br>G <sup>g</sup> | Schedule H <sup>h</sup> | Schedule I <sup>i</sup> | Schedule J <sup>j</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Double-Blind Perio | d | | | | | | | | | | |
| Baseline | 1 | ≤1 | ≤1 | ≤1 | ≤1 | ≤1 | | ≤1 | ≤ 1 | ≤1 | ≤ 1 |
| Week 2 | 15 | >1*- 21 | | | | | | | >1*-21 | >1*-49 | |
| Week 4 | 29 | 22-42 | | | | >1*-56 | >1*-56 | >1*-42 | 22 - 56 | | >1*-98 |
| Week 8 | 57 | 43-70 | | | | | | 43 - 70 | | | |
| Week 12 | 85 | 71-98 | >1*-126 | >1*-126 | | 57 - 126 | 57 - 126 | 71 - 98 | 57 - 98 | 50 - 126 | |
| Week 16 | 113 | 99-126 | | | | | | 99 - 126 | 99 - 140 | | |
| Week 20 | 141 | 127-154 | | | | | | 127 - 154 | | | |
| Week 24 | 169 | 155-196 | 127 - 224 | 127 - 266 | | 127 - 224 | 127 - 224 | 155 - 196 | 141 - 266 | 127 - 266 | ≥ 99 |
| Week 32 | 225 | 197-252 | | | | | | 197 - 252 | | | |
| Week 40 | 281 | 253-322 | 225 - 322 | | | 225 - 322 | 225 - 322 | 253 - 322 | | | |
| Week 52 | 365 | ≥323 | ≥ 323 | ≥ 267 | >1* | ≥ 323 | ≥ 323 | ≥ 323 | ≥ 267 | ≥ 267 | |

a Includes temperature, heart rate, blood pressure, GCA clinical assessments (including disease flare), CRP, ESR

b Includes weight, glucocorticoid toxicity index (excluding bone density assessment)

c Includes physician global assessments (MD-VAS), patient reported outcomes and antibodies to sarilumab/ADA

d Includes bone density assessment, ANA

e Includes hematology: hemoglobin, hematocrit, red blood cell (RBC) count and morphology (if RBC count is abnormal), white blood cell (WBC) differential, platelet count, absolute neutrophil count (ANC) and chemistry: sodium, potassium, calcium, chloride, bicarbonate, total protein, creatinine and clearance, blood urea nitrogen (BUN), uric acid, lactate dehydrogenase (LDH), phosphate, albumin, ALT (SGPT), AST (SGOT), alkaline phosphatase (ALP), total bilirubin, conjugated bilirubin, and unconjugated bilirubin

f Includes HbA1c, fasting glucose, fasting lipids: triglycerides (TG), total cholesterol, HDL, LDL

g Includes urine pregnancy test

h Includes serum sarilumab

i Includes biomarkers-IL-6 and sIL-6R

j Includes immune cell phenotyping (whole blood)

<sup>\*</sup> Includes value measured on day 1 but after the first IMP dose

For PK and ADA, the follow-up (i.e., 6-week post-treatment) measurement will be defined based on the sample collected at the follow-up visit (ie, Visit 13). The rests of PK and ADA measurements will be mapped to each visit using the visit window defined in Table 9.

# Appendix I Baseline glucocorticoid toxicity

Approach to calculating the Baseline glucocorticoid toxicity score: Toxicities assigned weighted scores from the Composite Index to establish a baseline glucocorticoid toxicity score

| Toxicity Domain | | Points |
|---|---|---|
| | BMI < 27 | 0 |
| Body Mass Index (BMI) | BMI > 27 but < 30 | 21 |
| | BMI > 30 | 36 |
| Glucose Metabolism | HgbA1c < 5.7 | 0 |
| | HgbA1c < 5.7 but on medication | 32 |
| | Hgb A1c > 5.7 | 32 |
| | HgbA1c > 5.7 and on medication | 44 |
| | Diabetic retinopathy, nephropathy, or neuropathy (count only one) | 44 |
| | LDL < target <sup>a</sup> | 0 |
| Lipid Metabolism | LDL < target <sup>a</sup> but on medications | 10 |
| | LDL > target <sup>a</sup> on no medications | 10 |
| | LDL > target <sup>a</sup> on treatment | 30 |
| | Normal BMD or no known history of osteoporosis | 0 |
| | Osteoporosis | 29 |
| Bone/Tendon | Insufficiency fracture secondary to osteoporosis | |
| | Osteonecrosis | 29 |
| | Tendon rupture while on corticosteroid | 29 |
| | No myopathy | 0 |
| Glucocorticoid | Minor glucocorticoid myopathy | 9 |
| Myopathy | Moderate glucocorticoid myopathy | 63 |
| | Severe glucocorticoid myopathy | 63 |
| | No skin toxicity | 0 |
| a1 : | Minor skin toxicity (one or more than one minor skin item) | 8 |
| Skin | Moderate skin toxicity (one or more than one moderate skin item) | 26 |
| | Severe skin toxicity (one or more than one moderate skin item) | 26 |
| | No neuropsychiatric toxicity | 0 |
| Neuropsychiatric | Minor (one or more than one minor NP item: insomnia, mania, depression, cognitive) | |
| | Moderate (one or more than one moderate NP item: insomnia, mania, depression, cognitive) | 74 |
| | Severe (one or more than one severe NP item: insomnia, mania, depression, cognitive) | |
| | Psychosis | 74 |
| | Glucocorticoid-induced violence | 74 |
| | No GTI-relevant infections within the pre-baseline GTI interval of the | 0 |
| Infection | Oral or vaginal candidiasis or non-complicated zoster ( <grade3) gti="" interval="" of="" pre-baseline="" study<="" td="" the="" within=""><td>19</td></grade3)> | 19 |

| | Grade 3 or Grade 4 infection within the pre-baseline GTI interval of the study | 93 |
|---|---|---|
| | Increased IOP | 33 |
| Ocular | Posterior subcapsular cataract | 33 |
| | Central serous retinopathy | 33 |
| Gastrointestinal | GI perf absence of NSAIDs | 33 |
| | PUD without H. pylori | 33 |
| Endocrine | Adrenal insufficiency | 33 |

a Target range of <70 mg/dL will be used for LDL domain.

# Signature Page efc15068-16-1-9-sap

| Approve & eSign |
|-----------------|
| Approve & eSign |